CLINICAL TRIAL: NCT00565812
Title: A Long-Term, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Radiographic Study To Investigate The Safety And Efficacy Of Orally Administered SD-6010 In Subjects With Symptomatic Osteoarthritis Of The Knee
Brief Title: A Long-Term, Placebo-Controlled X-Ray Study Investigating the Safety and Efficacy of SD-6010 in Subjects With Osteoarthritis of the Knee
Acronym: ITIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A6171016; 2007-001457-26 (EudraCT Number); ITIC (Other: Alias Study Number)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Results first posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Osteoarthritis
Keywords: knee Osteoarthritis Disease Modifying Osteoarthritis Drug
MeSH Terms: conditions — Osteoarthritis | interventions — cindunistat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 200 mg (Active Comparator): High dose active comparator
  Interventions: Drug: SD-6010
- 50 mg (Active Comparator): Low dose active comparator
  Interventions: Drug: SD-6010
- Placebo (Placebo Comparator): Placebo comparator to be used for control purposes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SD-6010 — 200 mg tablets once a day for 2 years
  Arms: 200 mg
Drug: SD-6010 — 50 mg tablets once a day for 2 years
  Arms: 50 mg
Drug: Placebo — Placebo tablets once a day for 2 years
  Arms: Placebo

SUMMARY:
The objective of this 2-year study is to evaluate the safety, tolerability and disease modifying efficacy of SD 6010, an inhibitor of inducible nitric oxide synthase (iNOS), in overweight and obese subjects with knee osteoarthritis. The efficacy of SD-6010 will be evaluated by radiography using joint space narrowing in the medial tibiofemoral compartment of the study knee as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged >= 40 years with a BMI >= 25 and <= 40 kg/m2
* In the past, has been diagnosed with knee OA
* Radiographic evidence of OA in the study knee

Exclusion Criteria:

* A diagnosis of any other rheumatic disease
* Current conditions in the study knee that would confound efficacy
* Selected, traditional clinical safety and laboratory parameters

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1457 (Actual)
Dates: Start 2007-11; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (181):
- United States (118):
  - Brookwood Internists, P.C., Birmingham, Alabama
  - Greystone Medical Center, Birmingham, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Pivotal Research Centers, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Martin Bowen Hefley Orthopedics, Little Rock, Arkansas
  - Teton Research, LLC, Little Rock, Arkansas
  - Med Center, Carmichael, California
  - College Hospital Costa Mesa, Costa Mesa, California
  - NeuroNetwork Trials, Costa Mesa, California
  - Med Investigations, Inc., Fair Oaks, California
  - Sierra Clinical Research, Roseville, California
  - University of California Davis Health System, Sacramento, California
  - University of California Davis, Sacramento, California
  - Scripps Clinic-Clinical Research, San Diego, California
  - Plaza Medical Imaging, Santa Ana, California
  - Denver Internal Medicine Group, Denver, Colorado
  - Mountain View Clinical Research, Inc., Denver, Colorado
  - New West Physicians Clinical Research, Golden, Colorado
  - Advanced Radiology Consultants, Fairfield, Connecticut
  - Advanced Radiology Consultants, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Southeastern Arthritis Center, Gainesville, Florida
  - Southeastern Imaging & Diagnostics, Gainesville, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research Institute, Gainesville, Florida
  - Jacksonville Center for Clincal Research, Jacksonville, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Marin E. Hale, M.D., P.A., Plantation, Florida
  - Sabiha Khan, M.D., Plantation, Florida
  - Kanner, Mendelson, Shteinman, LLC, West Palm Beach, Florida
  - Radiant Research, West Palm Beach, Florida
  - Rheumatology and Endocrinology Specialists of the Palm Beaches, P.A., West Palm Beach, Florida
  - North Georgia Clinical Research, Marietta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Preventive Medicine, Chicago, Illinois
  - Rehabilitation Institue of Chicago, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Illinois Bone and Joint Institute, LLC, Morton Grove, Illinois
  - The Arthritis Center, Springfield, Illinois
  - NorthShore University HealthSystem, Vernon Hills, Illinois
  - Ronald Keith Stegemoller, American Health Network, Avon, Indiana
  - Floyd Memorial Hospital, New Albany, Indiana
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Family Medicine East, Chartered/Radiology, Wichita, Kansas
  - Office of Manoj Kohli, M.D., Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - TFD Research, LLC, Shreveport, Louisiana
  - Rheumatology Associates, Portland, Maine
  - The Center for Rheumatology and Bone Research, Rockville, Maryland
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Miray Medical Center, Brockton, Massachusetts
  - Phase III Clinical Research, Fall River, Massachusetts
  - Fall River Clinical Research, Fall River, Massachusetts
  - HCI Metromedic Walk-In, New Bedford, Massachusetts
  - MedVadis Research Corporation, Wellesley Hills, Massachusetts
  - Fallon Clinic, Inc. (Drug Shipment), Worcester, Massachusetts
  - Fallon Clinic, Inc., Worcester, Massachusetts
  - Cadillac Clinical Research, LLC, located at Great Lakes Family Care, Cadillac, Michigan
  - Arthritis and Osteoporosis Treatment and Research Center, Flowood, Mississippi
  - Planters Clinic, Port Gibson, Mississippi
  - North Mississippi Medical Center, Inc., Tupelo, Mississippi
  - Mercy Medical Group/Woodlake Research, Clarkson Valley, Missouri
  - Dynamic Clinical Research, Inc., Kansas City, Missouri
  - Joan Prouty Moore, MD, Kansas City, Missouri
  - Orthopaedic and Occupational Medicine, Kansas City, Missouri
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - Office of Michael Mall, M.D., Las Vegas, Nevada
  - Nevada Imaging Centers, Las Vegas, Nevada
  - Office of Danka Michaels, MD, Las Vegas, Nevada
  - Office of Stephen H. Miller, MD, Las Vegas, Nevada
  - Regional Clinical Research, Inc., Endwell, New York
  - NYU Hospital for Joint Diseases, New York, New York
  - VirtualScopics, Inc., Rochester, New York
  - Crouse Medical Practice, PLLC d/b/a Internist Associates of Central New York, Syracuse, New York
  - Kernodle Clinic Inc., Burlington, North Carolina
  - Southeastern Radiology, Greensboro, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Research Institute of the Carolinas, PLLC, Mooresville, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - Carolina Arthritis Associates, PA, Wilmington, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Internal Medicine Associates, Fargo, North Dakota
  - Lillestol Research, LLC, Fargo, North Dakota
  - Advantage Diagnostics, Beachwood, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - Optimed Research, LLC, Columbus, Ohio
  - Lake Health Lyndhurst Clinic, Lyndhurst, Ohio
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - BioImaging Technologies, Inc., Newtown, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rheumatology Associates, Charleston, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Parkway Medical Group, Fayetteville, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - D. Matthew Sellers MD PC, Knoxville, Tennessee
  - Southwind Medical Specialists, Memphis, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Radiant Research San Antonio Northeast, San Antonio, Texas
  - South Texas Radiology Imaging Center, San Antonio, Texas
  - Oakwell Clinical Research, LLC, San Antonio, Texas
  - Pivotal Research Centers, Midvale, Utah
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research, Incorporated, Richmond, Virginia
  - Advanced Pain Management, Virginia Beach, Virginia
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
- Argentina (5):
  - OMI - Organización Médica de Investigación, Buenos Aires
  - Saint Dennis Medical Group S.A., Buenos Aires
  - Investigaciones Reumatológicas y Osteológicas S.R.L., Buenos Aires
  - Instituto Médico Especializado (IME), Buenos Aires
  - IMAI Research, Buenos Aires
- Menzies Research Institute, Hobart, Tasmania, Australia
- Belgium (2):
  - Cliniques Universitaires St Luc, Brussels
  - Universitair Ziekenhuis Gasthuisberg / Rheumatology, Leuven
- Canada (4):
  - Rheumatology Research Associates Ltd., Edmonton, Alberta
  - Nexus Clinic Research, St. John's, Newfoundland and Labrador
  - The Arthritis Program Research Group Inc., Newmarket, Ontario
  - Centre de Rhumatologie St-Louis, Sainte-Foy, Quebec
- Czechia (14):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno-Židenice
  - MEDIPONT Plus, s.r.o., České Budějovice
  - MEDIPONT, s.r.o., České Budějovice
  - ARTMEDI UPD s r.o., Hostivice
  - Nemocnice Na Frantisku s poliklinikou, Prague
  - Revmatologicky ustav, Prague
  - Centrum pro zdravotnicke zabezpeceni sportovni reprezentace, Prague
  - Ustredni vojenska nemocnice Praha, Prague
  - MSI - Muskuloskeletalni institut, Prague
  - DC Mediscan, Praha 11 - Chodov
  - MediCentrum Praha, a.s., Praha 11 - Chodov
  - Nemocnice Atlas, a.s., Zlín
  - PV-Medical s.r.o., Zlín
- Germany (5):
  - Praxis fuer Orthopaedie, Chirotherapie und Akupunktur, Bad Hersfeld
  - Praxis fuer Orthopaedie, Berlin
  - Klinische Forschung Berlin-Buch, Berlin
  - Praxis Dr. Thomas Jung, Deggingen
  - Klinische Forschung Schwerin, Schwerin
- Hungary (7):
  - Orszagos Gerincgyogyaszati Kozpont, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - Heves Megyei Onkormanyzat Markhot Ferenc Korhaz, Eger
  - Bekes Megyei Kepviselo-testulet Pandy Kalman Korhaz, Reumatologia, Gyula
  - Selye Janos Korhaz, Reumatologiai Szakrendelo, Komárom
  - MAV Korhaz es Rendelointezet, Szolnok
  - Veszprem Megyei Onkormanyzat Csolnoky Ferenc Korhaz-Rendelointezet, Veszprém
- Italy (3):
  - Azienda Sanitaria Genovese, Ospedale La Colletta, Dipartimento Apparato Locomotore, Arenzano
  - Presidio Ospedaliero Augusto Murri, Reparto di Reumatologia, Jesi (Ancona)
  - Ospedale Luigi Sacco, Azienda Ospedaliera Polo Universitario Unita' Operativa di Reumatologia, Milan
- Peru (8):
  - Clínica San Felipe, Lima, Lima Province
  - Hospital Nacional "Edgardo Rebagliati Martins" - Essalud, Lima, Lima Province
  - Instituto Peruano del Hueso y la Articulación SAC., Lima, Lima Province
  - Hospital Maria Auxiliadora, Lima, Lima Province
  - Centro Medico Corpac, Lima, Lima Province
  - Centro Empresarial - Altavista Polo 4, Santiago de Surco, Lima region
  - Instituto de Ginecologia y Reproducción & Cirugia Minimamente Invasiva, Santiago de Surco, Lima region
  - Hospital Nacional "Alberto Sabogal Sologuren" - Essalud, Callao, Provincia Constitucional del Callao
- Poland (3):
  - NSZOZ "MEDICUS II" S.C. Irena Klimczak, Malgorzata Klimczak, Jerzy Klimczak, Cieszyn
  - "SYNEXUS SCM" Sp. z o.o., Wroclaw
  - Katedra i Klinika Ortopedii i Traumatologii Narzadu Ruchu, Wroclaw
- Russia (5):
  - Russian State Medical University, Moscow Faculty, City Clinical Hospital #4, Moscow
  - Institute of Rheumatology, Moscow
  - City Alexandrovskaya Hospital, Saint Petersburg
  - L.G. Sokolov Clinical Hospital #122 of Federal Medical-Biology Agency of Russia, Central Polyclinic, Saint Petersburg
  - Research Institute of Traumatology and Orthopedy Named After R. R. Vredena, Saint Petersburg
- Slovakia (3):
  - V. Interna klinika FN a LF UK, Bratislava
  - Ivan Ujvari, Bratislava
  - Narodny ustav reumatickych chorob, Piešťany
- Spain (3):
  - Hospital Ntra. Sra. de La Esperanza, Santiago de Compostela, A Coruña
  - Hospital General Universitario de Guadalajara, Guadalajara, Guadalajara
  - Hospital Nuestra Señora de Valme, Seville, Sevilla

REFERENCES:
- [Derived] Hellio le Graverand MP, Clemmer RS, Redifer P, Brunell RM, Hayes CW, Brandt KD, Abramson SB, Manning PT, Miller CG, Vignon E. A 2-year randomised, double-blind, placebo-controlled, multicentre study of oral selective iNOS inhibitor, cindunistat (SD-6010), in patients with symptomatic osteoarthritis of the knee. Ann Rheum Dis. 2013 Feb;72(2):187-95. doi: 10.1136/annrheumdis-2012-202239. Epub 2012 Nov 10. PMID 23144445
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6171016&StudyName=A%20Long-Term%2C%20Placebo-Controlled%20X-Ray%20Study%20Investigating%20the%20Safety%20and%20Efficacy%20of%20SD-6010%20in%20Subjects%20with%20Osteoarthritis%20of%20the%20Knee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5077 participants were screened in the study, out of which only 1457 participants were randomized.
Groups:
- SD-6010 50 Milligram (mg): Participants with symptomatic osteoarthritis (OA) of knee, received 50 mg tablet of SD-6010 orally, once daily for 24 months.
- SD-6010 200 mg: Participants with symptomatic OA of knee, received 200 mg tablet of SD-6010 orally, once daily for 24 months.
- Placebo: Participants with symptomatic OA of knee, received placebo matched to SD-6010 orally, once daily for 24 months.
Period: Overall Study
Arm/Group | SD-6010 50 Milligram (mg) | SD-6010 200 mg | Placebo
Started | 485 | 486 | 486
Completed | 341 | 351 | 356
Not Completed | 144 | 135 | 130
Not completed — Death | 2 | 1 | 3
Not completed — Did not Meet Entrance Criteria | 1 | 0 | 1
Not completed — Lost to Follow-up | 10 | 8 | 8
Not completed — Withdrawal by Subject | 58 | 47 | 48
Not completed — Work Schedule | 5 | 3 | 1
Not completed — Protocol Violation | 2 | 6 | 4
Not completed — Adverse Event | 41 | 54 | 40
Not completed — Jury Duty | 1 | 0 | 0
Not completed — Relocated Out of Area | 5 | 8 | 9
Not completed — Sponsor Decision | 1 | 5 | 1
Not completed — Domestic Reasons | 7 | 1 | 3
Not completed — Research Site Closure | 6 | 1 | 8
Not completed — Surgical Intervention | 0 | 1 | 2
Not completed — Low Compliance | 1 | 0 | 1
Not completed — Follow-up Visit Not Completed | 2 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants randomized to the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | SD-6010 50 Milligram (mg) | SD-6010 200 mg | Placebo | Total
Number analyzed (Participants) | 485 | 486 | 486 | 1457
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (8.7) | 60.8 (8.6) | 61.3 (9.1) | 61.0 (8.8)
Gender [Count of Participants; unit: Participants]
  Female | 383 | 367 | 364 | 1114
  Male | 102 | 119 | 122 | 343

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression of Joint Space Narrowing
Description: Rate of progression of joint space narrowing (JSN) was defined as narrowing in joint space width (JSW) over the course of the study. It was measured radiographically in the medial tibiofemoral of knee of participants with OA. The slope reported in millimeter per year (mm/year) over a 2 year period was used to assess the rate of progression of JSN. Negative values indicating a worsening of osteoarthritis.
Time Frame: Baseline up to Month 24
Population: FAS included all participants randomized to the study. Here, 'number of participants analyzed' (N) signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/year
Groups:
- SD-0610 50 Milligram (mg): Participants with symptomatic osteoarthritis (OA) of knee, received 50 mg tablet of SD-6010 orally, once daily for 24 months.
- SD-0610 200 mg: Participants with symptomatic OA of knee, received 200 mg tablet of SD-6010 orally, once daily for 24 months.
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 422 | 428 | 434
mm/year | -0.101 (0.346) [-0.128 to -0.078] | -0.125 (0.298) [-0.134 to -0.085] | -0.109 (0.261) [-0.139 to -0.091]
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Slopes, 95 percent confidence interval (CI), P-values: Random coefficients mixed-effects model for repeated measures (MMRM) with random intercept and slope for each participant,fixed effects for treatment group,time (years),treatment group*time interaction,(collapsed)Kellgren and Lawrence Grades (KLG), KLG*time interaction,geographic region,gender,age,body mass index with unstructured covariance matrix for random effects. Statistical hypothesis used Hochberg procedure with 2-sided alpha =0.0499; Test type: Superiority or Other; p = 0.508770, Mixed Models Analysis; Difference in Slopes = 0.012, 95% CI 2-sided [-0.023 to 0.046], Standard Error of Mean 0.018
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; Slopes, 95 percent CI, P-values: MMRM with random intercept and slope for each participant, fixed effects for treatment group, time (years), treatment group*time interaction, (collapsed) KLG, KLG*time interaction, geographic region, gender, age, body mass index with unstructured covariance matrix for random effects. Statistical hypothesis used Hochberg procedure with 2-sided alpha=0.0499; Test type: Superiority or Other; p = 0.754074, Mixed Models Analysis; Difference in Slopes = 0.005, 95% CI 2-sided [-0.029 to 0.040], Standard Error of Mean 0.017

2. Primary Outcome: Rate of Progression of Joint Space Narrowing in Participants With Kellgren and Lawrence Grade Less Than or Equal to (<=) 2
Description: Rate of progression of JSN was defined as narrowing in joint space width over the course of the study. It was measured radiographically in the medial tibiofemoral of knee of participants with OA. The slope reported in mm/year over a 2 year period was used to assess the rate of progression of JSN. KLG system was a method of classifying the severity of knee OA using five grades (0 [no severity] to 4 [maximum severity], higher grade indicating worse knee function). Negative values of slope indicating a worsening of osteoarthritis.
Time Frame: Baseline up to Month 24
Population: FAS included all participants randomized to the study. Here, 'N' signifies participants with KLG <=2 and evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 184 | 172 | 194
mm/year | -0.061 (0.335) [-0.087 to -0.023] | -0.069 (0.254) [-0.088 to -0.022] | -0.075 (0.221) [-0.108 to -0.047]
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Slopes, 95 percent CI and P-values were obtained from a random coefficients MMRM with random intercept and slope for each participant, and fixed effects for treatment group, time (years), a treatment group*time (years) interaction, geographic region, gender, age, and body mass index with an unstructured covariance matrix for the random effects; Test type: Superiority or Other; p = 0.312, Mixed Models Analysis; Difference in slopes = 0.023, 95% CI 2-sided [-0.022 to 0.067], Standard Error of Mean 0.023
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.327, Mixed Models Analysis; Difference in slopes = 0.022, 95% CI 2-sided [-0.022 to 0.067], Standard Error of Mean 0.023

3. Primary Outcome: Rate of Progression of Joint Space Narrowing in Participants With Kellgren and Lawrence Grade Equal to (=) 3
Description: as for outcome 2
Time Frame: Baseline up to Month 24
Population: FAS included all participants randomized to the study. Here, 'N' signifies participants with KLG =3 and evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mm/year
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 238 | 256 | 240
mm/year | -0.133 (0.352) [-0.176 to -0.104] | -0.162 (0.319) [-0.185 to -0.117] | -0.136 (0.286) [-0.179 to -0.109]
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.881, Mixed Models Analysis; Difference in slopes = 0.004, 95% CI 2-sided [-0.046 to 0.054], Standard Error of Mean 0.026
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.780, Mixed Models Analysis; Difference in slopes = -0.007, 95% CI 2-sided [-0.056 to 0.042], Standard Error of Mean 0.025

4. Secondary Outcome: Change From Baseline in Western Ontario and MacMaster Osteoarthritis Index (WOMAC) Composite Index Score at Month 3, 6, 12, 18 and 24
Description: The WOMAC was a self-administered, disease-specific instrument which probed clinically important, participant relevant symptoms in the areas of pain, stiffness, and physical function in participants with OA of the knee. The WOMAC composite index was the sum of 24 individual questions regarding subscales of pain, stiffness and physical function (for each item score range: 0 [minimum] to 4 [maximum], higher score indicating worse knee condition). Total score was sum of the 3 subscale scores, giving a possible overall score range of 0 (minimum) to 96 (maximum). Higher score indicating the worse level of pain, stiffness and physical function.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: FAS included all participants randomized to the study. Here, 'n' signifies participants evaluable for this outcome measure at given time points for each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 481) | 39.07 (18.85) | 37.29 (17.98) | 38.45 (18.91)
  Change at Month 3 (n =449, 450, 455) | -5.35 (14.73) | -5.08 (13.14) | -5.50 (13.59)
  Change at Month 6 (n =424, 426, 433) | -7.20 (15.99) | -5.84 (15.15) | -7.07 (15.62)
  Change at Month 12 (n =370, 388, 397) | -9.17 (18.19) | -9.25 (15.82) | -9.84 (15.75)
  Change at Month 18 (n =344, 361, 357) | -9.91 (17.98) | -8.35 (16.87) | -8.82 (18.00)
  Change at Month 24 (n =336, 339, 349) | -10.85 (18.49) | -10.98 (17.62) | -10.49 (17.26)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 3; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.639, Mixed Models Analysis; LS mean difference = 0.40, 95% CI 2-sided [-1.26 to 2.05], Standard Error of Mean 0.84
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; Month 3; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.957, Mixed Models Analysis; LS mean difference = 0.05, 95% CI 2-sided [-1.61 to 1.70], Standard Error of Mean 0.84
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 6; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.893, Mixed Models Analysis; LS mean difference = 0.13, 95% CI 2-sided [-1.76 to 2.01], Standard Error of Mean 0.96
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.365, Mixed Models Analysis; LS mean difference = 0.87, 95% CI 2-sided [-1.01 to 2.76], Standard Error of Mean 0.96
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 12; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.678, Mixed Models Analysis; LS mean difference = 0.44, 95% CI 2-sided [-1.63 to 2.51], Standard Error of Mean 1.05
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.902, Mixed Models Analysis; LS mean difference = -0.13, 95% CI 2-sided [-2.18 to 1.93], Standard Error of Mean 1.05
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 18; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.577, Mixed Models Analysis; LS mean difference = -0.64, 95% CI 2-sided [-2.89 to 1.61], Standard Error of Mean 1.15
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.980, Mixed Models Analysis; LS mean difference = -0.03, 95% CI 2-sided [-2.26 to 2.21], Standard Error of Mean 1.14
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 24; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.950, Mixed Models Analysis; LS mean difference = -0.07, 95% CI 2-sided [-2.37 to 2.23], Standard Error of Mean 1.17
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.292, Mixed Models Analysis; LS mean difference = -1.23, 95% CI 2-sided [-3.53 to 1.06], Standard Error of Mean 1.17

5. Secondary Outcome: Change From Baseline in Western Ontario and MacMaster Osteoarthritis Index Pain Subscale Score at Month 3, 6, 12, 18 and 24
Description: The WOMAC pain subscale was comprised of 5 questions regarding the amount of pain experienced due to OA in the study knee. The WOMAC pain subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse pain. An overall subscale score range of 0 (minimum) to 20 (maximum), with higher scores indicating more pain.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =482, 484, 483) | 7.96 (3.94) | 7.44 (3.87) | 7.59 (4.03)
  Change at Month 3 (n =451, 453, 458) | -1.32 (3.41) | -1.23 (3.19) | -1.25 (3.15)
  Change at Month 6 (n =426, 429, 435) | -1.73 (3.73) | -1.42 (3.58) | -1.59 (3.45)
  Change at Month 12 (n =372, 389, 398) | -2.17 (4.25) | -2.10 (3.66) | -2.08 (3.47)
  Change at Month 18 (n =347, 363, 359) | -2.24 (4.16) | -2.00 (3.93) | -1.86 (3.88)
  Change at Month 24 (n =337, 342, 351) | -2.48 (4.02) | -2.23 (4.16) | -2.19 (3.79)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 3; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group* visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.683, Mixed Models Analysis; LS mean difference = 0.08, 95% CI 2-sided [-0.30 to 0.46], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; Month 3; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.853, Mixed Models Analysis; LS mean difference = -0.04, 95% CI 2-sided [-0.42 to 0.35], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 6; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group* visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis; LS mean difference = 0.02, 95% CI 2-sided [-0.41 to 0.44], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; Month 6; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.648, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-0.32 to 0.52], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.916, Mixed Models Analysis; LS mean difference = -0.02, 95% CI 2-sided [-0.49 to 0.44], Standard Error of Mean 0.24
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.528, Mixed Models Analysis; LS mean difference = -0.15, 95% CI 2-sided [-0.60 to 0.31], Standard Error of Mean 0.23
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 18; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.365, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-0.73 to 0.27], Standard Error of Mean 0.25
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 7]; Test type: Superiority or Other; p = 0.328, Mixed Models Analysis; LS mean difference = -0.25, 95% CI 2-sided [-0.74 to 0.25], Standard Error of Mean 0.25
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.540, Mixed Models Analysis; LS mean difference = -0.16, 95% CI 2-sided [-0.66 to 0.35], Standard Error of Mean 0.26
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 9]; Test type: Superiority or Other; p = 0.423, Mixed Models Analysis; LS mean difference = -0.21, 95% CI 2-sided [-0.71 to 0.30], Standard Error of Mean 0.26

6. Secondary Outcome: Change From Baseline in Western Ontario and MacMaster Osteoarthritis Index Pain Stiffness Subscale Score at Month 3, 6, 12, 18 and 24
Description: Stiffness was defined as a sensation of decreased ease in which the participant moved the knee with OA. The WOMAC stiffness subscale was comprised of 2 questions regarding the degree of stiffness experienced in the study knee. The WOMAC stiffness subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse stiffness. An overall score range of 0 (minimum) to 8 (maximum), with higher scores indicating more stiffness.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 484, 482) | 3.48 (1.80) | 3.33 (1.78) | 3.44 (1.77)
  Change at Month 3 (n =449, 455, 456) | -0.52 (1.67) | -0.51 (1.58) | -0.51 (1.58)
  Change at Month 6 (n =425, 429, 434) | -0.67 (1.70) | -0.56 (1.78) | -0.62 (1.73)
  Change at Month 12 (n =371, 389, 397) | -0.89 (1.89) | -0.79 (1.83) | -0.95 (1.78)
  Change at Month 18 (n =346, 363, 358) | -0.88 (1.86) | -0.87 (1.88) | -0.82 (1.82)
  Change at Month 24 (n =336, 342, 349) | -0.94 (1.95) | -1.10 (1.95) | -0.95 (1.92)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.904, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-0.17 to 0.20], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.582, Mixed Models Analysis; LS mean difference = -0.05, 95% CI 2-sided [-0.24 to 0.13], Standard Error of Mean 0.09
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 6; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.818, Mixed Models Analysis; LS mean difference = -0.02, 95% CI 2-sided [-0.22 to 0.18], Standard Error of Mean 0.10
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; Month 6; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group x visit interaction, (collapsed) KLG, a (collapsed) KLG x visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.988, Mixed Models Analysis; LS mean difference = -0.00, 95% CI 2-sided [-0.20 to 0.20], Standard Error of Mean 0.10
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 12; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.857, Mixed Models Analysis; LS mean difference = 0.02, 95% CI 2-sided [-0.20 to 0.24], Standard Error of Mean 0.11
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; Month 12; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.658, Mixed Models Analysis; LS mean difference = 0.05, 95% CI 2-sided [-0.17 to 0.27], Standard Error of Mean 0.11
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.612, Mixed Models Analysis; LS mean difference = -0.06, 95% CI 2-sided [-0.28 to 0.17], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.391, Mixed Models Analysis; LS mean difference = -0.10, 95% CI 2-sided [-0.32 to 0.13], Standard Error of Mean 0.11
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 24; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value,geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 1.000, Mixed Models Analysis; LS mean difference = -0.00, 95% CI 2-sided [-0.24 to 0.24], Standard Error of Mean 0.12
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; Month 24; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis; LS mean difference = -0.21, 95% CI 2-sided [-0.45 to 0.03], Standard Error of Mean 0.12

7. Secondary Outcome: Change From Baseline in Western Ontario and MacMaster Osteoarthritis Index Physical Function Subscale Score at Month 3, 6, 12, 18 and 24
Description: The WOMAC physical function subscale referred to the participant's ability to move around and perform usual activities of daily living. The WOMAC physical function subscale was comprised of 17 questions regarding the degree of difficulty experienced due to OA in the study knee. The WOMAC physical function subscale score for each question ranged from 0 (minimum) to 4 (maximum), higher scores signified worse physical function. An overall score range of 0 (minimum) to 68 (maximum), with higher scores indicating worse physical function.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 482) | 27.63 (13.88) | 26.49 (13.18) | 27.39 (13.81)
  Change at Month 3 (n =449, 452, 456) | -3.50 (10.77) | -3.24 (9.71) | -3.72 (9.99)
  Change at Month 6 (n =424, 426, 434) | -4.78 (11.73) | -3.86 (10.81) | -4.82 (11.43)
  Change at Month 12 (n =370, 388, 398) | -6.09 (13.21) | -6.37 (11.34) | -6.79 (11.55)
  Change at Month 18 (n =344, 361, 358) | -6.74 (12.95) | -5.49 (12.05) | -6.12 (13.22)
  Change at Month 24 (n =336, 339, 350) | -7.42 (13.47) | -7.65 (12.37) | -7.35 (12.54)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.586, Mixed Models Analysis; LS mean difference = 0.34, 95% CI 2-sided [-0.88 to 1.55], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.789, Mixed Models Analysis; LS mean difference = 0.17, 95% CI 2-sided [-1.05 to 1.38], Standard Error of Mean 0.62
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.821, Mixed Models Analysis; LS mean difference = 0.16, 95% CI 2-sided [-1.21 to 1.52], Standard Error of Mean 0.69
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.294, Mixed Models Analysis; LS mean difference = 0.73, 95% CI 2-sided [-0.63 to 2.09], Standard Error of Mean 0.69
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.532, Mixed Models Analysis; LS mean difference = 0.48, 95% CI 2-sided [-1.02 to 1.97], Standard Error of Mean 0.76
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis; LS mean difference = -0.06, 95% CI 2-sided [-1.55 to 1.43], Standard Error of Mean 0.76
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.680, Mixed Models Analysis; LS mean difference = -0.34, 95% CI 2-sided [-1.97 to 1.29], Standard Error of Mean 0.83
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.730, Mixed Models Analysis; LS mean difference = 0.28, 95% CI 2-sided [-1.33 to 1.90], Standard Error of Mean 0.82
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.901, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-1.55 to 1.76], Standard Error of Mean 0.84
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.333, Mixed Models Analysis; LS mean difference = -0.81, 95% CI 2-sided [-2.45 to 0.83], Standard Error of Mean 0.84

8. Secondary Outcome: Change From Baseline in Patient Assessment of Arthritic Pain Visual Analog Scale (VAS) Score at Month 3, 6, 12, 18 and 24
Description: Pain VAS was a self-administered instrument, a 100 millimeter (mm) line marked by participant. Intensity of pain range (over past week): 0 (mm) =no pain to 100 (mm) =worst possible pain. Higher score indicating severe pain.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
mm
  Baseline (n =478, 479, 482) | 40.19 (24.77) | 37.59 (24.26) | 39.37 (23.91)
  Change at Month 3 (n =446, 448, 455) | -7.21 (25.49) | -7.02 (23.45) | -9.12 (21.72)
  Change at Month 6 (n =422, 424, 435) | -10.13 (24.91) | -7.92 (24.90) | -10.17 (24.07)
  Change at Month 12 (n =370, 384, 396) | -11.75 (30.38) | -10.98 (25.28) | -12.97 (24.26)
  Change at Month 18 (n =342, 360, 360) | -13.99 (26.78) | -11.17 (25.60) | -12.86 (26.47)
  Change at Month 24 (n =333, 338, 348) | -14.59 (28.36) | -13.36 (25.69) | -13.29 (23.97)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.086, Mixed Models Analysis; LS mean difference = 2.34, 95% CI 2-sided [-0.33 to 5.01], Standard Error of Mean 1.36
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.415, Mixed Models Analysis; LS mean difference = 1.11, 95% CI 2-sided [-1.56 to 3.78], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.569, Mixed Models Analysis; LS mean difference = 0.80, 95% CI 2-sided [-1.97 to 3.57], Standard Error of Mean 1.41
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.374, Mixed Models Analysis; LS mean difference = 1.26, 95% CI 2-sided [-1.51 to 4.02], Standard Error of Mean 1.41
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.288, Mixed Models Analysis; LS mean difference = 1.63, 95% CI 2-sided [-1.38 to 4.64], Standard Error of Mean 1.53
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.440, Mixed Models Analysis; LS mean difference = 1.18, 95% CI 2-sided [-1.81 to 4.17], Standard Error of Mean 1.52
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.896, Mixed Models Analysis; LS mean difference = -0.21, 95% CI 2-sided [-3.30 to 2.88], Standard Error of Mean 1.58
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.464, Mixed Models Analysis; LS mean difference = 1.14, 95% CI 2-sided [-1.92 to 4.20], Standard Error of Mean 1.56
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.901, Mixed Models Analysis; LS mean difference = -0.20, 95% CI 2-sided [-3.27 to 2.88], Standard Error of Mean 1.57
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 9]; Test type: Superiority or Other; p = 0.800, Mixed Models Analysis; LS mean difference = -0.39, 95% CI 2-sided [-3.45 to 2.66], Standard Error of Mean 1.56

9. Secondary Outcome: Change From Baseline in Patient Global Assessment of Arthritic Condition Score at Month 3, 6, 12, 18 and 24
Description: Participants answered: "Considering all the ways your arthritis affects you, how are you feeling today?" Participants responded by using the scale ranging from 1 (minimum) to 5 (maximum), where 1 =very good, 2 =good, 3 =fair, 4 =poor and 5 =very poor. Higher scores indicating worse condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 483) | 2.684 (0.904) | 2.610 (0.883) | 2.634 (0.883)
  Change at Month 3 (n =449, 452, 455) | -0.232 (0.909) | -0.230 (0.816) | -0.202 (0.787)
  Change at Month 6 (n =424, 427, 435) | -0.337 (0.876) | -0.319 (0.857) | -0.260 (0.879)
  Change at Month 12 (n =368, 385, 397) | -0.405 (0.908) | -0.371 (0.930) | -0.370 (0.848)
  Change at Month 18 (n =344, 361, 358) | -0.442 (0.979) | -0.418 (0.934) | -0.388 (0.903)
  Change at Month 24 (n =335, 340, 351) | -0.513 (0.950) | -0.488 (0.939) | -0.473 (0.934)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.984, Mixed Models Analysis; LS mean difference = 0.001, 95% CI 2-sided [-0.093 to 0.095], Standard Error of Mean 0.048
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.330, Mixed Models Analysis; LS mean difference = -0.046, 95% CI 2-sided [-0.140 to 0.047], Standard Error of Mean 0.048
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.308, Mixed Models Analysis; LS mean difference = -0.050, 95% CI 2-sided [-0.146 to 0.046], Standard Error of Mean 0.049
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis; LS mean difference = -0.083, 95% CI 2-sided [-0.180 to 0.013], Standard Error of Mean 0.049
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.508, Mixed Models Analysis; LS mean difference = -0.035, 95% CI 2-sided [-0.137 to 0.068], Standard Error of Mean 0.052
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.490, Mixed Models Analysis; LS mean difference = -0.036, 95% CI 2-sided [-0.137 to 0.066], Standard Error of Mean 0.052
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.739, Mixed Models Analysis; LS mean difference = -0.019, 95% CI 2-sided [-0.132 to 0.094], Standard Error of Mean 0.057
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis; LS mean difference = -0.050, 95% CI 2-sided [-0.162 to 0.061], Standard Error of Mean 0.057
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.883, Mixed Models Analysis; LS mean difference = -0.008, 95% CI 2-sided [-0.121 to 0.104], Standard Error of Mean 0.057
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.690, Mixed Models Analysis; LS mean difference = -0.023, 95% CI 2-sided [-0.135 to 0.089], Standard Error of Mean 0.057

10. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Arthritic Condition Score at Month 3, 6, 12, 18 and 24
Description: Physician assessed the overall impact of arthritis on the participant's daily life. Participant's condition was rated by the physician using the scale ranging from 1 (minimum) to 5 (maximum), where 1= very good, 2= good, 3= fair, 4= poor and 5= very poor. Higher scores indicating worse condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =480, 483, 480) | 2.785 (0.679) | 2.834 (0.689) | 2.831 (0.655)
  Change at Month 3 (n =449, 448, 453) | -0.379 (0.782) | -0.422 (0.756) | -0.415 (0.764)
  Change at Month 6 (n =420, 426, 431) | -0.443 (0.823) | -0.561 (0.841) | -0.452 (0.791)
  Change at Month 12 (n =367, 386, 396) | -0.548 (0.873) | -0.627 (0.859) | -0.535 (0.828)
  Change at Month 18 (n =342, 359, 355) | -0.602 (0.906) | -0.643 (0.833) | -0.628 (0.862)
  Change at Month 24 (n = 331, 340, 349) | -0.656 (0.906) | -0.662 (0.879) | -0.711 (0.867)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.849, Mixed Models Analysis; LS mean difference = 0.008, 95% CI 2-sided [-0.078 to 0.095], Standard Error of Mean 0.044
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.837, Mixed Models Analysis; LS mean difference = -0.009, 95% CI 2-sided [-0.096 to 0.078], Standard Error of Mean 0.044
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.776, Mixed Models Analysis; LS mean difference = -0.013, 95% CI 2-sided [-0.105 to 0.078], Standard Error of Mean 0.047
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis; LS mean difference = -0.100, 95% CI 2-sided [-0.191 to -0.008], Standard Error of Mean 0.047
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.201, Mixed Models Analysis; LS mean difference = -0.064, 95% CI 2-sided [-0.163 to 0.034], Standard Error of Mean 0.050
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; LS mean difference = -0.103, 95% CI 2-sided [-0.201 to -0.006], Standard Error of Mean 0.050
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.848, Mixed Models Analysis; LS mean difference = -0.010, 95% CI 2-sided [-0.114 to 0.094], Standard Error of Mean 0.053
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.714, Mixed Models Analysis; LS mean difference = -0.019, 95% CI 2-sided [-0.122 to 0.084], Standard Error of Mean 0.052
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.652, Mixed Models Analysis; LS mean difference = 0.025, 95% CI 2-sided [-0.082 to 0.131], Standard Error of Mean 0.054
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.700, Mixed Models Analysis; LS mean difference = 0.021, 95% CI 2-sided [-0.085 to 0.127], Standard Error of Mean 0.054

11. Secondary Outcome: Change From Baseline in Pain After a 50-foot Walk Using Pain Visual Analog Scale Score at Month 3, 6, 12, 18 and 24
Description: The pain VAS following a 50 foot walk was a single-item, self-administered instrument. Participants were asked to assess the pain due to OA in their study knee after a 50-foot walk. Participants responded on a VAS scale ranging from 0 (no pain) to 100 (severe pain). Higher scores indicating more pain.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =480, 483, 482) | 38.03 (26.39) | 35.13 (26.10) | 38.00 (25.73)
  Change at Month 3 (n =446, 453, 456) | -5.78 (25.30) | -5.71 (23.20) | -7.45 (23.15)
  Change at Month 6 (n =424, 428, 436) | -8.13 (25.86) | -7.17 (25.42) | -8.78 (25.67)
  Change at Month 12 (n =370, 382, 397) | -11.32 (27.42) | -10.07 (25.22) | -11.91 (24.04)
  Change at Month 18 (n = 345, 360, 357) | -11.17 (27.51) | -8.91 (27.12) | -11.86 (26.04)
  Change at Month 24 (n =336, 340, 351) | -12.31 (27.61) | -12.86 (26.73) | -13.77 (24.53)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.220, Mixed Models Analysis; LS mean difference = 1.68, 95% CI 2-sided [-1.00 to 4.36], Standard Error of Mean 1.37
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.997, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-2.67 to 2.68], Standard Error of Mean 1.36
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.613, Mixed Models Analysis; LS mean difference = 0.73, 95% CI 2-sided [-2.09 to 3.55], Standard Error of Mean 1.44
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.964, Mixed Models Analysis; LS mean difference = 0.06, 95% CI 2-sided [-2.75 to 2.88], Standard Error of Mean 1.44
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.872, Mixed Models Analysis; LS mean difference = 0.24, 95% CI 2-sided [-2.69 to 3.17], Standard Error of Mean 1.49
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.947, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-2.81 to 3.01], Standard Error of Mean 1.48
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.927, Mixed Models Analysis; LS mean difference = 0.15, 95% CI 2-sided [-3.03 to 3.33], Standard Error of Mean 1.62
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.547, Mixed Models Analysis; LS mean difference = 0.97, 95% CI 2-sided [-2.18 to 4.12], Standard Error of Mean 1.61
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.304, Mixed Models Analysis; LS mean difference = 1.62, 95% CI 2-sided [-1.47 to 4.71], Standard Error of Mean 1.58
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.679, Mixed Models Analysis; LS mean difference = -0.65, 95% CI 2-sided [-3.73 to 2.43], Standard Error of Mean 1.57

12. Secondary Outcome: Change From Baseline in Osteoarthritis Pain Assessment Tool-Knee Joint Total Score at Month 3, 6, 12, 18 and 24
Description: The OA pain and assessment tool-knee joint is also known as the intermittent and constant osteoarthritis pain (ICOAP) scale. The OA pain assessment tool-knee joint was an 11-item scale, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst health condition. The total score was calculated by adding the 11 items and rescaled to a 0 (minimum) to 100 (maximum) scale, where higher scores indicating worse health.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: FAS included all participants randomized to the study. Here, 'n' signifies participants evaluated for this outcome measure at given time points for each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =479, 480, 481) | 39.35 (23.06) | 36.55 (21.78) | 38.79 (22.29)
  Change at Month 3 (n =448, 450, 449) | -7.00 (19.95) | -6.68 (17.77) | -7.08 (18.15)
  Change at Month 6 (n =422, 422, 430) | -9.09 (21.43) | -7.74 (19.36) | -8.27 (19.68)
  Change at Month 12 (n = 365, 384, 397) | -13.00 (21.93) | -10.84 (20.58) | -12.26 (20.24)
  Change at Month 18 (n =342, 359, 359) | -12.71 (22.64) | -9.59 (21.26) | -11.23 (22.13)
  Change at Month 24 (n =330, 340, 349) | -13.02 (22.30) | -12.87 (21.53) | -13.79 (21.81)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.738, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [-1.80 to 2.55], Standard Error of Mean 1.11
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.632, Mixed Models Analysis; LS mean difference = -0.53, 95% CI 2-sided [-2.70 to 1.64], Standard Error of Mean 1.11
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.736, Mixed Models Analysis; LS mean difference = -0.41, 95% CI 2-sided [-2.77 to 1.96], Standard Error of Mean 1.21
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.811, Mixed Models Analysis; LS mean difference = -0.29, 95% CI 2-sided [-2.66 to 2.08], Standard Error of Mean 1.21
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.335, Mixed Models Analysis; LS mean difference = -1.22, 95% CI 2-sided [-3.71 to 1.26], Standard Error of Mean 1.27
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.966, Mixed Models Analysis; LS mean difference = -0.05, 95% CI 2-sided [-2.52 to 2.41], Standard Error of Mean 1.26
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.299, Mixed Models Analysis; LS mean difference = -1.44, 95% CI 2-sided [-4.16 to 1.28], Standard Error of Mean 1.38
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.925, Mixed Models Analysis; LS mean difference = 0.13, 95% CI 2-sided [-2.56 to 2.82], Standard Error of Mean 1.37
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.676, Mixed Models Analysis; LS mean difference = 0.58, 95% CI 2-sided [-2.14 to 3.30], Standard Error of Mean 1.39
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.732, Mixed Models Analysis; LS mean difference = -0.47, 95% CI 2-sided [-3.18 to 2.23], Standard Error of Mean 1.38

13. Secondary Outcome: Change From Baseline in Osteoarthritis Pain Assessment Tool-Knee Joint Constant Pain Subscale Score at Month 3, 6, 12, 18 and 24
Description: The OA pain assessment tool-knee joint constant pain subscale was a 5 item scale, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst health condition. Overall subscale score was calculated by adding the 5 items and rescaled to a 0 (minimum) to 100 (maximum) scale, where higher scores indicating worse constant pain.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =479, 481, 484) | 35.25 (24.83) | 33.01 (24.09) | 35.21 (24.45)
  Change at Month 3 (n =448, 452, 454) | -6.61 (21.64) | -6.41 (19.44) | -6.55 (19.92)
  Change at Month 6 (n =423, 426, 434) | -7.88 (23.11) | -7.47 (21.05) | -8.25 (20.55)
  Change at Month 12 (n = 367, 384, 399) | -11.78 (23.21) | -10.83 (21.94) | -11.75 (21.85)
  Change at Month 18 (n = 343, 360, 360) | -11.63 (23.68) | -9.88 (22.01) | -10.62 (23.82)
  Change at Month 24 (n = 330, 340, 350) | -11.59 (23.68) | -12.51 (23.17) | -13.15 (23.37)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.911, Mixed Models Analysis; LS mean difference = 0.13, 95% CI 2-sided [-2.22 to 2.49], Standard Error of Mean 1.20
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.500, Mixed Models Analysis; LS mean difference = -0.81, 95% CI 2-sided [-3.16 to 1.54], Standard Error of Mean 1.20
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.596, Mixed Models Analysis; LS mean difference = 0.67, 95% CI 2-sided [-1.81 to 3.15], Standard Error of Mean 1.26
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.979, Mixed Models Analysis; LS mean difference = -0.03, 95% CI 2-sided [-2.51 to 2.44], Standard Error of Mean 1.26
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis; LS mean difference = -0.59, 95% CI 2-sided [-3.20 to 2.03], Standard Error of Mean 1.33
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.823, Mixed Models Analysis; LS mean difference = -0.30, 95% CI 2-sided [-2.89 to 2.30], Standard Error of Mean 1.32
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.387, Mixed Models Analysis; LS mean difference = -1.24, 95% CI 2-sided [-4.04 to 1.57], Standard Error of Mean 1.43
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.737, Mixed Models Analysis; LS mean difference = -0.48, 95% CI 2-sided [-3.25 to 2.30], Standard Error of Mean 1.42
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.443, Mixed Models Analysis; LS mean difference = 1.12, 95% CI 2-sided [-1.73 to 3.97], Standard Error of Mean 1.45
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.585, Mixed Models Analysis; LS mean difference = -0.79, 95% CI 2-sided [-3.62 to 2.04], Standard Error of Mean 1.44

14. Secondary Outcome: Change From Baseline in Osteoarthritis Pain Assessment Tool-Knee Joint Intermittent Pain Subscale Score at Month 3, 6, 12, 18 and 24
Description: The OA pain assessment tool-knee joint intermittent pain subscale score a 6 item scale, with each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst health condition. Overall subscale score was calculated by adding the 6 items and rescaled to a 0 (minimum) to 100 (maximum) scale, where higher scores indicating worse intermittent pain.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =479, 480, 481) | 42.76 (22.85) | 39.44 (21.46) | 41.73 (22.10)
  Change at Month 3 (n =448, 450, 450) | -7.32 (20.68) | -6.93 (18.95) | -7.48 (19.28)
  Change at Month 6 (n =422, 422, 430) | -10.18 (22.28) | -7.96 (20.34) | -8.31 (21.44)
  Change at Month 12 (n =365, 385, 397) | -14.15 (22.93) | -10.93 (21.86) | -12.54 (21.64)
  Change at Month 18 (n =342, 359, 359) | -13.56 (23.72) | -9.45 (23.07) | -11.69 (23.02)
  Change at Month 24 (n =330, 340, 349) | -14.20 (23.11) | -13.17 (22.74) | -14.27 (22.66)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.613, Mixed Models Analysis; LS mean difference = 0.58, 95% CI 2-sided [-1.68 to 2.85], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.670, Mixed Models Analysis; LS mean difference = -0.49, 95% CI 2-sided [-2.76 to 1.78], Standard Error of Mean 1.16
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.296, Mixed Models Analysis; LS mean difference = -1.33, 95% CI 2-sided [-3.82 to 1.16], Standard Error of Mean 1.27
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.604, Mixed Models Analysis; LS mean difference = -0.66, 95% CI 2-sided [-3.15 to 1.83], Standard Error of Mean 1.27
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.163, Mixed Models Analysis; LS mean difference = -1.86, 95% CI 2-sided [-4.46 to 0.75], Standard Error of Mean 1.33
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.939, Mixed Models Analysis; LS mean difference = -0.10, 95% CI 2-sided [-2.69 to 2.48], Standard Error of Mean 1.32
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.233, Mixed Models Analysis; LS mean difference = -1.74, 95% CI 2-sided [-4.61 to 1.12], Standard Error of Mean 1.46
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.720, Mixed Models Analysis; LS mean difference = 0.52, 95% CI 2-sided [-2.32 to 3.36], Standard Error of Mean 1.45
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.993, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-2.82 to 2.85], Standard Error of Mean 1.45
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.794, Mixed Models Analysis; LS mean difference = -0.38, 95% CI 2-sided [-3.19 to 2.44], Standard Error of Mean 1.44

15. Secondary Outcome: Change From Baseline in Osteoarthritis Research Society International (OARSI) Knee Function Survey Score at Month 3, 6, 12, 18 and 24
Description: The OARSI knee function survey was an 11-item scale with each item scored 0 (minimum) to 4 (maximum), where 4 indicated worst health condition. The total score was the sum of the 11 items and ranged from 0 (minimum) to 44 (maximum), where higher scores indicating worse health condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =382, 376, 391) | 22.19 (8.96) | 21.49 (8.59) | 21.80 (8.92)
  Change at Month 3 (n = 309, 304, 315) | -2.20 (7.70) | -2.24 (6.57) | -2.99 (7.12)
  Change at Month 6 (n =270, 283, 294) | -3.24 (8.42) | -3.29 (7.80) | -3.53 (8.26)
  Change at Month 12 (n =240, 263, 266) | -4.57 (8.65) | -4.35 (7.76) | -4.46 (7.99)
  Change at Month 18 (n =225, 239, 243) | -5.14 (9.37) | -4.61 (8.56) | -4.93 (9.22)
  Change at Month 24(n = 227, 224, 237) | -5.31 (9.40) | -5.13 (8.36) | -5.62 (9.28)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.069, Mixed Models Analysis; LS mean difference = 0.97, 95% CI 2-sided [-0.07 to 2.02], Standard Error of Mean 0.53
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.335, Mixed Models Analysis; LS mean difference = 0.52, 95% CI 2-sided [-0.53 to 1.57], Standard Error of Mean 0.54
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis; LS mean difference = 0.89, 95% CI 2-sided [-0.33 to 2.11], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.672, Mixed Models Analysis; LS mean difference = 0.26, 95% CI 2-sided [-0.95 to 1.47], Standard Error of Mean 0.62
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.765, Mixed Models Analysis; LS mean difference = 0.19, 95% CI 2-sided [-1.05 to 1.43], Standard Error of Mean 0.63
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.675, Mixed Models Analysis; LS mean difference = 0.26, 95% CI 2-sided [-0.96 to 1.49], Standard Error of Mean 0.62
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.560, Mixed Models Analysis; LS mean difference = 0.42, 95% CI 2-sided [-1.00 to 1.84], Standard Error of Mean 0.72
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.433, Mixed Models Analysis; LS mean difference = 0.56, 95% CI 2-sided [-0.84 to 1.97], Standard Error of Mean 0.72
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.318, Mixed Models Analysis; LS mean difference = 0.73, 95% CI 2-sided [-0.70 to 2.16], Standard Error of Mean 0.73
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.303, Mixed Models Analysis; LS mean difference = 0.75, 95% CI 2-sided [-0.68 to 2.18], Standard Error of Mean 0.73

16. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS) Score at Month 3, 6, 12, 18 and 24
Description: The KOOS-PS was used to rate participant's opinions about the difficulties they experienced with activity due to problems with their knee. It was a 7-item scale, each item scored from 0 (minimum) to 4 (maximum), where 4 indicated worst health condition. Total score was calculated by adding the responses to 7 items and rescaled to a 0 (minimum) to 100 (maximum) scale, where higher scores indicating worse health condition.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =432, 423, 428) | 42.75 (14.69) | 41.82 (13.85) | 42.60 (14.76)
  Change at Month 3 (n =376, 363, 370) | -3.50 (12.68) | -4.31 (11.38) | -5.23 (11.47)
  Change at Month 6 (n =336, 335, 348) | -5.42 (13.70) | -5.41 (13.93) | -6.03 (14.02)
  Change at Month 12 (n =288, 315, 320) | -7.01 (14.60) | -7.67 (13.26) | -7.32 (13.52)
  Change at Month 18 (n =284, 284, 280) | -8.10 (16.00) | -7.44 (14.09) | -7.47 (15.00)
  Change at Month 24 (n =272, 272, 278) | -8.49 (16.06) | -9.01 (14.74) | -9.60 (15.48)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 3; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLGU*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis; LS mean difference = 1.67, 95% CI 2-sided [0.08 to 3.26], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p = 0.395, Mixed Models Analysis; LS mean difference = 0.70, 95% CI 2-sided [-0.91 to 2.30], Standard Error of Mean 0.82
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.160, Mixed Models Analysis; LS mean difference = 1.36, 95% CI 2-sided [-0.54 to 3.25], Standard Error of Mean 0.96
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.638, Mixed Models Analysis; LS mean difference = 0.46, 95% CI 2-sided [-1.44 to 2.35], Standard Error of Mean 0.97
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.537, Mixed Models Analysis; LS mean difference = 0.61, 95% CI 2-sided [-1.32 to 2.54], Standard Error of Mean 0.98
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; Month 12; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*(visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.988, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-1.90 to 1.93], Standard Error of Mean 0.98
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.962, Mixed Models Analysis; LS mean difference = 0.05, 95% CI 2-sided [-2.12 to 2.22], Standard Error of Mean 1.11
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.856, Mixed Models Analysis; LS mean difference = 0.20, 95% CI 2-sided [-1.97 to 2.37], Standard Error of Mean 1.11
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.237, Mixed Models Analysis; LS mean difference = 1.36, 95% CI 2-sided [-0.90 to 3.63], Standard Error of Mean 1.15
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.475, Mixed Models Analysis; LS mean difference = 0.82, 95% CI 2-sided [-1.44 to 3.09], Standard Error of Mean 1.15

17. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Functioning Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 16.18 (minimum) to 57.11 (maximum), with higher scores indicating better physical functioning.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 485) | 35.67 (9.74) | 36.84 (9.42) | 36.32 (9.15)
  Change at Month 12 (n =368, 381, 397) | 2.59 (8.80) | 2.41 (8.66) | 2.55 (8.84)
  Change at Month 24 (n =332, 341, 352) | 3.53 (9.50) | 3.23 (9.66) | 3.51 (9.54)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.938, Mixed Models Analysis; LS mean difference = 0.04, 95% CI 2-sided [-1.07 to 1.16], Standard Error of Mean 0.57
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.906, Mixed Models Analysis; LS mean difference = 0.07, 95% CI 2-sided [-1.04 to 1.17], Standard Error of Mean 0.56
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.726, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-1.50 to 1.04], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.681, Mixed Models Analysis; LS mean difference = -0.26, 95% CI 2-sided [-1.52 to 1.00], Standard Error of Mean 0.64

18. Secondary Outcome: Change From Baseline in Short Form-36 Role - Physical Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 18.45 (minimum) to 56.62 (maximum), with higher scores indicating better role-physical.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 485) | 39.99 (9.85) | 40.37 (9.73) | 40.14 (10.03)
  Change at Month 12 (n =368, 381, 397) | 2.06 (9.55) | 2.35 (8.75) | 2.22 (8.85)
  Change at Month 24 (n =333, 341, 352) | 2.44 (9.53) | 2.44 (9.34) | 2.70 (9.35)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.900, Mixed Models Analysis; LS mean difference = 0.07, 95% CI 2-sided [-1.07 to 1.21], Standard Error of Mean 0.58
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.528, Mixed Models Analysis; LS mean difference = 0.36, 95% CI 2-sided [-0.77 to 1.50], Standard Error of Mean 0.58
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.647, Mixed Models Analysis; LS mean difference = -0.29, 95% CI 2-sided [-1.51 to 0.94], Standard Error of Mean 0.62
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.841, Mixed Models Analysis; LS mean difference = -0.12, 95% CI 2-sided [-1.34 to 1.09], Standard Error of Mean 0.62

19. Secondary Outcome: Change From Baseline in Short Form-36 Bodily Pain Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 19.23 (minimum) to 60.88 (maximum), with higher scores indicating lower bodily pain.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 485) | 38.81 (8.63) | 39.77 (8.34) | 38.90 (8.22)
  Change at Month 12 (n =368, 381, 397) | 4.07 (9.64) | 3.72 (8.32) | 4.06 (8.97)
  Change at Month 24 (n =332, 341, 352) | 4.25 (9.54) | 4.65 (9.90) | 4.46 (9.44)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.587, Mixed Models Analysis; LS mean difference = 0.32, 95% CI 2-sided [-0.84 to 1.48], Standard Error of Mean 0.59
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.687, Mixed Models Analysis; LS mean difference = 0.24, 95% CI 2-sided [-0.91 to 1.38], Standard Error of Mean 0.58
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.677, Mixed Models Analysis; LS mean difference = -0.27, 95% CI 2-sided [-1.56 to 1.01], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.469, Mixed Models Analysis; LS mean difference = 0.47, 95% CI 2-sided [-0.80 to 1.74], Standard Error of Mean 0.65

20. Secondary Outcome: Change From Baseline in Short Form-36 General Health Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 16.75 (minimum) to 63.72 (maximum), with higher scores indicating better general health.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 481, 484) | 44.77 (10.15) | 46.49 (9.79) | 45.19 (9.63)
  Change at Month 12 (n =367, 381, 395) | 1.33 (7.52) | 1.10 (7.64) | 1.20 (6.93)
  Change at Month 24 (n =331, 341, 352) | 1.13 (8.43) | 0.40 (7.76) | 1.25 (7.77)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.632, Mixed Models Analysis; LS mean difference = 0.23, 95% CI 2-sided [-0.71 to 1.17], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.308, Mixed Models Analysis; LS mean difference = 0.49, 95% CI 2-sided [-0.45 to 1.42], Standard Error of Mean 0.48
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.615, Mixed Models Analysis; LS mean difference = -0.27, 95% CI 2-sided [-1.33 to 0.79], Standard Error of Mean 0.54
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.425, Mixed Models Analysis; LS mean difference = -0.43, 95% CI 2-sided [-1.48 to 0.62], Standard Error of Mean 0.53

21. Secondary Outcome: Change From Baseline in Short Form-36 Vitality Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 22.02 (minimum) to 69.92 (maximum), with higher scores indicating better vitality.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 481, 484) | 47.57 (9.44) | 49.00 (9.20) | 48.08 (9.53)
  Change at Month 12 (n =368, 381, 396) | 1.52 (8.51) | 0.48 (8.04) | 1.04 (8.22)
  Change at Month 24 (n =332, 340, 351) | 1.53 (8.71) | 0.78 (8.62) | 1.42 (8.70)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.214, Mixed Models Analysis; LS mean difference = 0.67, 95% CI 2-sided [-0.39 to 1.72], Standard Error of Mean 0.54
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.980, Mixed Models Analysis; LS mean difference = -0.01, 95% CI 2-sided [-1.06 to 1.03], Standard Error of Mean 0.53
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.575, Mixed Models Analysis; LS mean difference = 0.33, 95% CI 2-sided [-0.83 to 1.49], Standard Error of Mean 0.59
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.986, Mixed Models Analysis; LS mean difference = -0.01, 95% CI 2-sided [-1.16 to 1.14], Standard Error of Mean 0.59

22. Secondary Outcome: Change From Baseline in Short Form-36 Social Functioning Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 13.38 (minimum) to 56.40 (maximum), with higher scores indicating better social functioning.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 485) | 45.15 (11.06) | 46.23 (10.19) | 45.64 (10.36)
  Change at Month 12 (n =368, 381, 397) | 1.11 (10.28) | -0.28 (9.16) | -0.15 (9.74)
  Change at Month 24 (n =333, 341, 352) | 1.31 (10.62) | 0.88 (10.15) | 0.12 (10.03)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.030, Mixed Models Analysis; LS mean difference = 1.33, 95% CI 2-sided [0.13 to 2.52], Standard Error of Mean 0.61
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.480, Mixed Models Analysis; LS mean difference = 0.43, 95% CI 2-sided [-0.76 to 1.61], Standard Error of Mean 0.60
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.132, Mixed Models Analysis; LS mean difference = 1.01, 95% CI 2-sided [-0.30 to 2.32], Standard Error of Mean 0.67
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.117, Mixed Models Analysis; LS mean difference = 1.04, 95% CI 2-sided [-0.26 to 2.34], Standard Error of Mean 0.66

23. Secondary Outcome: Change From Baseline in Short Form-36 Role-Emotional Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 10.25 (minimum) to 55.68 (maximum), with higher scores indicating better role-emotional.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 482, 485) | 43.73 (12.79) | 43.27 (12.09) | 43.37 (12.35)
  Change at Month 12 (n =368, 381, 396) | 0.05 (12.06) | -0.18 (10.55) | -0.25 (11.47)
  Change at Month 24 (n =333, 341, 352) | -0.28 (12.77) | 0.60 (11.69) | 0.32 (11.98)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.133, Mixed Models Analysis; LS mean difference = 1.06, 95% CI 2-sided [-0.32 to 2.44], Standard Error of Mean 0.71
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.524, Mixed Models Analysis; LS mean difference = 0.44, 95% CI 2-sided [-0.93 to 1.82], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.743, Mixed Models Analysis; LS mean difference = 0.26, 95% CI 2-sided [-1.27 to 1.78], Standard Error of Mean 0.78
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.310, Mixed Models Analysis; LS mean difference = 0.78, 95% CI 2-sided [-0.73 to 2.30], Standard Error of Mean 0.77

24. Secondary Outcome: Change From Baseline in Short Form-36 Mental Health Domain Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 8.02 (minimum) to 63.43 (maximum), with higher scores indicating better mental health.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 481, 484) | 47.01 (10.80) | 47.70 (10.73) | 47.26 (11.15)
  Change at Month 12 (n =368, 381, 396) | 0.95 (10.08) | 0.19 (9.10) | -0.31 (9.50)
  Change at Month 24 (n =332, 340, 351) | 1.12 (10.26) | 0.26 (10.01) | -0.01 (9.81)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.058, Mixed Models Analysis; LS mean difference = 1.17, 95% CI 2-sided [-0.04 to 2.38], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.213, Mixed Models Analysis; LS mean difference = 0.76, 95% CI 2-sided [-0.44 to 1.96], Standard Error of Mean 0.61
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.143, Mixed Models Analysis; LS mean difference = 0.98, 95% CI 2-sided [-0.33 to 2.30], Standard Error of Mean 0.67
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.450, Mixed Models Analysis; LS mean difference = 0.50, 95% CI 2-sided [-0.80 to 1.81], Standard Error of Mean 0.67

25. Secondary Outcome: Change From Baseline in Short Form-36 Physical Health Component Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 22.88 (minimum) to 58.69 (maximum), with higher scores indicating better physical health.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 480, 483) | 37.38 (8.84) | 38.69 (8.35) | 37.84 (8.46)
  Change at Month 12 (n =367, 381, 395) | 3.26 (7.98) | 3.31 (7.69) | 3.58 (7.87)
  Change at Month 24 (n =329, 340, 351) | 3.77 (8.48) | 3.66 (8.32) | 4.18 (8.48)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.701, Mixed Models Analysis; LS Mean Difference = -0.20, 95% CI 2-sided [-1.19 to 0.80], Standard Error of Mean 0.51
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.764, Mixed Models Analysis; LS Mean Difference = 0.15, 95% CI 2-sided [-0.84 to 1.14], Standard Error of Mean 0.50
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.228, Mixed Models Analysis; LS Mean Difference = -0.68, 95% CI 2-sided [-1.80 to 0.43], Standard Error of Mean 0.57
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; Month 24; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit,a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.514, Mixed Models Analysis; LS mean difference = -0.37, 95% CI 2-sided [-1.47 to 0.74], Standard Error of Mean 0.56

26. Secondary Outcome: Change From Baseline in Short Form-36 Mental Health Component Score at Month 12 and 24
Description: The SF-36 was a participant administered scale assessing general quality of life. It consisted of self-administered 36-item questionnaire that measured 8 health domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. These 8 domains were also summarized as physical and mental component scores. The score for each domain and component score was the mean of the individual question scores, which were scaled from 0 (minimum) to 100 (maximum), where higher scores indicated highest level of health/functioning. Linear transformations were performed to transform scores and rescaled to a score range of 11.11 (minimum) to 61.67 (maximum), with higher scores indicating better mental health.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =481, 480, 483) | 49.65 (11.79) | 49.97 (11.11) | 49.65 (11.62)
  Change at Month 12 (n =367, 381, 395) | -0.13 (10.64) | -1.17 (9.48) | -1.27 (9.65)
  Change at Month 24 (n =329, 340, 351) | -0.41 (11.24) | -0.70 (10.08) | -1.09 (10.18)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; LS mean difference = 1.42, 95% CI 2-sided [0.19 to 2.65], Standard Error of Mean 0.62
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 6]; Test type: Superiority or Other; p = 0.391, Mixed Models Analysis; LS mean difference = 0.53, 95% CI 2-sided [-0.68 to 1.75], Standard Error of Mean 0.62
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.142, Mixed Models Analysis; LS mean difference = 1.02, 95% CI 2-sided [-0.34 to 2.37], Standard Error of Mean 0.69
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 6, analysis 10]; Test type: Superiority or Other; p = 0.204, Mixed Models Analysis; LS mean difference = 0.87, 95% CI 2-sided [-0.47 to 2.21], Standard Error of Mean 0.68

27. Secondary Outcome: Number of Participants With EuroQoL-5D (EQ-5D) Mobility Domain Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health state profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. EQ-5D mobility domain score scale ranged from 1 (minimum) to 3 (maximum), where 1 =better health (no problem), 2 =moderate health (some problems) and 3 =worst health (confined to bed). Higher scores indicating worse health condition. Participants with EQ-5D mobility domain score were reported in this measure.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Baseline: No problem (n =481, 481, 485) | 132 | 135 | 163
  Baseline: Some problems (n =481, 481, 485) | 348 | 345 | 322
  Baseline: Confined to bed (n =481, 481, 485) | 1 | 1 | 0
  Month 12: No problem (n =371, 382, 399) | 174 | 186 | 178
  Month 12: Some problems (n =371, 382, 399) | 197 | 196 | 221
  Month 12: Confined to bed (n =371, 382, 399) | 0 | 0 | 0
  Month 24: No problem (n =334, 341, 353) | 167 | 161 | 178
  Month 24: Some problems (n =334, 341, 353) | 165 | 180 | 175
  Month 24: Confined to bed (n =334, 341, 353) | 2 | 0 | 0

28. Secondary Outcome: Number of Participants With EuroQoL-5D Self-Care Domain Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health state profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. EQ-5D self-care domain score scale ranged from 1 (minimum) to 3 (maximum), where 1 =better health (no problems with self-care), 2 =moderate health (some problems) and 3 =worst health (unable to wash or dress). Higher scores indicating worse health condition. Participants with EQ-5D self-care domain score were reported in this measure.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Baseline: No problem (n =480, 481, 485) | 383 | 387 | 386
  Baseline: Some problems (n =480, 481, 485) | 92 | 93 | 97
  Baseline: Unable to wash/dress (n =480, 481, 485) | 5 | 1 | 2
  Month 12: No problem (n =371, 382, 399) | 305 | 327 | 331
  Month 12: Some problems (n =371, 382, 399) | 66 | 51 | 67
  Month 12: Unable to wash/dress (n =371, 382, 399) | 0 | 4 | 1
  Month 24: No problem (n =334, 341, 352) | 280 | 286 | 299
  Month 24: Some problems (n =334, 341, 352) | 54 | 55 | 51
  Month 24: Unable to wash/dress (n =334, 341, 352) | 0 | 0 | 2

29. Secondary Outcome: Number of Participants With EuroQoL-5D Usual Activity Domain Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health state profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. EQ-5D usual activity domain score scale ranged from 1 (minimum) to 3 (maximum), where 1 =better health (no problems), 2 =moderate health (some problems) and 3 =worst health state (unable to perform usual activities). Higher scores indicating worse health condition. Participants with EQ-5D usual activity domain score were reported in this measure.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Baseline: No problem (n =481, 481, 485) | 186 | 185 | 190
  Baseline: Some problems (n =481, 481, 485) | 285 | 291 | 289
  Baseline: Unable to do activities(n=481,481,485) | 10 | 5 | 6
  Month 12: No problem (n =371, 382, 399) | 192 | 201 | 193
  Month 12: Some problems (n =371, 382, 399) | 176 | 180 | 204
  Month 12: Unable to do activities(n =371,382,399) | 3 | 1 | 2
  Month 24: No problem (n =334, 340, 352) | 187 | 186 | 205
  Month 24: Some problems (n =334, 340, 352) | 140 | 151 | 144
  Month 24: Unable to do activities(n =334,340,352) | 7 | 3 | 3

30. Secondary Outcome: Number of Participants With EuroQo-5D Pain and Discomfort Domain Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health state profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, anxiety and depression. EQ-5D pain and discomfort domain score scale ranged from 1 (minimum) to 3 (maximum), where 1 =better health (no pain and discomfort), 2 =moderate health (moderate pain and discomfort) and 3 =worst health state (extreme pain and discomfort). Higher scores indicated worse health condition. Participants with EQ-5D pain and discomfort domain score were reported in this measure.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Baseline: None (n =481, 481, 485) | 42 | 48 | 38
  Baseline: Moderate (n =481, 481, 485) | 383 | 391 | 403
  Baseline: Extreme (n =481, 481, 485) | 56 | 42 | 44
  Month 12: None (n =371, 382, 399) | 91 | 89 | 82
  Month 12: Moderate (n =371, 382, 399) | 259 | 280 | 293
  Month 12: Extreme (n =371, 382, 399) | 21 | 13 | 24
  Month 24: None (n =334, 341, 352) | 92 | 89 | 98
  Month 24: Moderate (n =334, 341, 352) | 226 | 232 | 240
  Month 24: Extreme (n =334, 341, 352) | 16 | 20 | 14

31. Secondary Outcome: Number of Participants With EuroQoL-5D Anxiety and Depression Domain Score
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life. Health state profile component assessed level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. EQ-5D anxiety and depression domain score scale ranged from 1 (minimum) to 3 (maximum), where 1 =better health (not anxious, depressed), 2 =moderate health (moderately anxious, depressed) and 3 =worst health (extremely anxious, depressed). Higher scores indicating worse health condition. Participants with EQ-5D anxiety and depression domain score were reported in this measure.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Baseline: None (n =481, 481, 485) | 297 | 306 | 303
  Baseline: Moderate (n =481, 481, 485) | 166 | 164 | 168
  Baseline: Extreme (n =481, 481, 485) | 18 | 11 | 14
  Month 12: None (n =371, 382, 399) | 251 | 256 | 261
  Month 12: Moderate (n =371, 382, 399) | 111 | 116 | 127
  Month12: Extreme (n =371, 382, 399) | 9 | 10 | 11
  Month 24: None (n =334, 341, 352) | 235 | 244 | 237
  Month 24: Moderate (n =334, 341, 352) | 93 | 89 | 109
  Month 24: Extreme (n =334, 341, 352) | 6 | 8 | 6

32. Secondary Outcome: EuroQoL-5D Visual Analog Scale Score
Description: The EQ-5D VAS score was a participant rated questionnaire to assess health-related quality of life in terms of a single index value. It was a visual analogue scale that ranged from 0 (minimum) to 100 (maximum), with higher scores indicating a better health condition.
Time Frame: Baseline, Month 12, 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
units on a scale
  Baseline (n =480, 479, 484) | 66.75 (21.52) | 68.59 (19.69) | 67.86 (19.36)
  Month 12 (n =369, 381, 399) | 72.34 (19.01) | 72.55 (19.48) | 70.58 (19.91)
  Month 24 (n =334, 341, 352) | 73.18 (19.64) | 73.95 (18.85) | 72.36 (19.36)

33. Secondary Outcome: Number of Participants With Increase in Total Analgesic Medication Use
Description: Increase in total analgesic medication use for OA in the study knee was a comparison back to baseline of an increased and sustained use of standard background and/or rescue medication for more than 28 days as measured at the Month 12 and 24 visits. Only medications for OA knee pain were considered.
Time Frame: Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Month 12 (n =372, 395, 408) | 21 | 29 | 24
  Month 24 (n =344, 353, 354) | 24 | 34 | 30
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 12; Odds ratio (OR), 95 percent CI and P-values were obtained from a logistic regression model, with treatment group, (collapsed) KLG, geographic region, and gender as factors, age and body mass index as covariates; Test type: Superiority or Other; p = 0.875, Regression, Logistic; Odds Ratio (OR) = 0.952, 95% CI 2-sided [0.516 to 1.756]
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; Month 12; Odds ratio, 95 percent CI and P-values were obtained from a logistic regression model, with treatment group, (collapsed) KLG, geographic region, and gender as factors, age and body mass index as covariates; Test type: Superiority or Other; p = 0.406, Regression, Logistic; Odds Ratio (OR) = 1.273, 95% CI 2-sided [0.721 to 2.247]
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Month 24; Odds ratio, 95 percent CI and P-values were obtained from a logistic regression model, with treatment group, (collapsed) KLG, geographic region, and gender as factors, age and body mass index as covariates; Test type: Superiority or Other; p = 0.406, Regression, Logistic; Odds Ratio (OR) = 0.787, 95% CI 2-sided [0.448 to 1.384]
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 33, analysis 3]; Test type: Superiority or Other; p = 0.591, Regression, Logistic; Odds Ratio (OR) = 1.154, 95% CI 2-sided [0.685 to 1.942]

34. Secondary Outcome: Number of Participants With Decrease in Total Analgesic Medication Use
Description: Decrease in total analgesic medication use for OA in the study knee was a comparison back to baseline of a decreased and irregular use of standard background and/or rescue medication for more than 28 days as measured at the Month 12 and 24 visits. Only medications for OA knee pain were considered.
Time Frame: Month 12, 24
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 485 | 486 | 486
participants
  Month 12 (n =372, 395, 408) | 29 | 38 | 43
  Month 24 (n =344, 353, 354) | 29 | 38 | 47
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.168, Regression, Logistic; Odds Ratio (OR) = 0.704, 95% CI 2-sided [0.428 to 1.160]
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 33, analysis 2]; Test type: Superiority or Other; p = 0.634, Regression, Logistic; Odds Ratio (OR) = 0.893, 95% CI 2-sided [0.560 to 1.423]
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 33, analysis 3]; Test type: Superiority or Other; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 0.583, 95% CI 2-sided [0.356 to 0.955]
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 33, analysis 3]; Test type: Superiority or Other; p = 0.276, Regression, Logistic; Odds Ratio (OR) = 0.774, 95% CI 2-sided [0.489 to 1.227]

35. Secondary Outcome: Patient Global Impression of Change Score
Description: Patient global impression of change was a participant-rated instrument that measured change in participant's overall status on a 7-point scale ranging from: 1 =very much improved, 2 =much improved, 3 =minimally improved, 4 =no change, 5 =minimally worse, 6 =much worse and 7 =very much worse. Higher scores indicating worse condition.
Time Frame: Month 24
Population: FAS included all participants randomized to the study. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 434 | 426 | 434
units on a scale | 2.97 (1.26) | 3.02 (1.34) | 3.00 (1.35)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; LS Mean, 95 percent CI and P-values were obtained from an analysis of covariance (ANCOVA) model, with treatment group, (collapsed) KLG, geographic region, and gender as factors and age and body mass index as covariates; Test type: Superiority or Other; p = 0.709, ANCOVA; LS mean difference = -0.03, 95% CI 2-sided [-0.21 to 0.14], Standard Error of Mean 0.09
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; LS-Mean, 95 percent CI and P-values were obtained from an ANCOVA model, with treatment group, (collapsed) KLG, geographic region, and gender as factors and age and body mass index as covariates; Test type: Superiority or Other; p = 0.798, ANCOVA; LS mean difference = 0.02, 95% CI 2-sided [-0.15 to 0.20], Standard Error of Mean 0.09

36. Secondary Outcome: Outcome Measures in Rheumatology-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: The OMERACT-OARSI responder index was used to determine whether participants may be considered responders to treatment. An OMERACT-OARSI responder was a participant who had a better response on the WOMAC pain subscale score, a better response on the WOMAC physical function subscale score or improvement on at least two of the three domains: WOMAC pain subscale score (overall score range of 0 [minimum] to 20 [maximum], higher scores indicating more pain), WOMAC physical function subscale score (overall score range of 0 [minimum] to 68 [maximum], higher scores indicating worse physical function) and patient global assessment of arthritic condition score (overall score range of 1 [minimum] to 5 [maximum], higher scores indicating worse condition). Number of participants who were OMERACT-OARSI responder were reported in this measure.
Time Frame: Month 24
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 468 | 469 | 470
participants | 222 | 226 | 219
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Odds ratio, 95 percent CI and P-values were obtained from a logistic regression model, with treatment group, (collapsed) KLG, geographic region, and gender as factors, baseline JSW, age and body mass index as covariates; Test type: Superiority or Other; p = 0.810, Regression, Logistic; Odds Ratio (OR) = 1.032, 95% CI 2-sided [0.797 to 1.337]
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 36, analysis 1]; Test type: Superiority or Other; p = 0.620, Regression, Logistic; Odds Ratio (OR) = 1.068, 95% CI 2-sided [0.824 to 1.383]

37. Secondary Outcome: Number of Participants With Joint Space Narrowing Progression
Description: JSN progressor was defined as a participant with a decrease in joint space width that was greater in magnitude than the smallest detectable difference (0.199 mm).
Time Frame: Month 24
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 419 | 423 | 429
participants | 136 | 153 | 165
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Odds ratio, 95 percent CI and P-values were obtained from a logistic regression model, with treatment group, (collapsed) KLG, geographic region, and gender as factors, age and body mass index as covariates; Test type: Superiority or Other; p = 0.047, Regression, Logistic; Odds Ratio (OR) = 0.745, 95% CI 2-sided [0.557 to 0.997]
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 37, analysis 1]; Test type: Superiority or Other; p = 0.317, Regression, Logistic; Odds Ratio (OR) = 0.864, 95% CI 2-sided [0.650 to 1.150]

38. Secondary Outcome: Number of Participants Applicable for Virtual Joint Replacement
Description: A virtual joint replacement candidate was defined as a participant whose last two WOMAC pain subscale scores (overall score range of 0 [minimum] to 20 [maximum], higher scores indicating more pain) were at least 8, last two WOMAC physical function subscale scores (overall score range of 0 [minimum] to 68 [maximum], higher scores indicating worse physical function) were at least 28 and was a joint space narrowing progressor (a participant with a decrease in JSW that was greater in magnitude than the smallest detectable difference =0.199 mm).
Time Frame: Month 24
Population: as for outcome 35
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 405 | 411 | 425
participants | 28 | 34 | 28
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 37, analysis 1]; Test type: Superiority or Other; p = 0.881, Regression, Logistic; Odds Ratio (OR) = 1.043, 95% CI 2-sided [0.602 to 1.806]
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 37, analysis 1]; Test type: Superiority or Other; p = 0.525, Regression, Logistic; Odds Ratio (OR) = 1.186, 95% CI 2-sided [0.701 to 2.009]

39. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 7-10 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. Adverse events included both serious and non-serious adverse events.
Time Frame: Baseline up to 7-10 days after last dose of study drug (Week 111)
Population: The safety analysis set included all participants in the FAS who received at least 1 dose of the randomized study medication.
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 482 | 485 | 485
participants
  Adverse events | 371 | 381 | 364
  Serious adverse events | 43 | 61 | 49

40. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Atrial (enlargement, fibrillation, premature beat), axis deviation, atrioventricular (accelerated conduction, first/second degree block), left anterior and posterior hemiblock, left atrial hypertrophy, left and right (complete/incomplete bundle branch block, ventricular hypertrophy), QRS (high/low voltage, nonspecific, prolongation greater than [>]140 milliseconds [msec]), junctional/paced rhythm, intraventricular conduction delay (>120 msec), early repolarization, ventricular premature contraction and beat, prolonged QTC, sinus (arrhythmia, bradycardia/tachycardia), supraventricular extra systole and premature beat, short PR syndrome. Abnormal Q-wave (>=30 msec), P-wave left/right atrial abnormality, T-wave flattened/inverted abnormality, U-wave abnormality, ST-T indeterminate abnormality, ST-T nonspecific changes, ST-T changes compatible with ischemia and pericarditis. ECG findings were judged by investigators for qualitative evaluation of abnormalities.
Time Frame: Baseline, Month 3, 6, 12, 18, 24
Population: The safety analysis set included all participants in the FAS who received at least 1 dose of the randomized study medication. Here, 'n' signifies participants evaluable for this outcome measure at given time points for each group.
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 482 | 485 | 485
participants
  Baseline (n =481, 484, 485) | 0 | 0 | 1
  Month 6 (n =414, 427, 427) | 3 | 0 | 1
  Month 12 (n =373 , 397, 403) | 4 | 1 | 2
  Month 18 (n =351, 366, 362) | 2 | 2 | 6
  Month 24 (n =338, 344, 351) | 3 | 1 | 6

41. Other Pre Specified Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Criteria for laboratory abnormalities: Hemoglobin (Hgb), hematocrit (hct), red blood cell(RBC) count: less than(<)0.8*lower limit of normal(LLN), platelet: <0.5*LLN or greater than (>)1.75*upper limit of normal (ULN), white blood cell (WBC): <0.6*LLN or >1.5*ULN, lymphocyte, neutrophil:<0.8*LLN or >1.2*ULN, basophil, eosinophil, monocyte:>1.2*ULN; total bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, gammaglutamyl transferase, alkaline phosphatase:> 3.0*ULN, total protein, albumin: <0.8*LLN or >1.2*ULN; blood urea nitrogen, creatinine:>1.3*ULN, uric acid >1.2*ULN; sodium <0.95*LLN or >1.05*ULN, potassium, chloride, calcium, magnesium, bicarbonate: <0.9*LLN or >1.1*ULN, phosphate <0.8*LLN or >1.2*ULN; glucose <0.6*LLN or >1.5*ULN, lipase >1.5*ULN; urine (specific gravity <1.003 or >1.030, pH <4.5 or >8, glucose, ketones, protein, blood/Hgb greater than or equal to [>=]1); pancreatic amylase >1.5*ULN.
Time Frame: Baseline up to Week 111
Population: The safety analysis set included all participants in the FAS who received at least 1 dose of the randomized study medication. Here, 'N' signifies participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 479 | 480 | 481
participants | 289 | 297 | 288

42. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 2, 4, 12, 24, 36, 48, 60, 72, 84 and 96
Description: Blood pressure (BP) was measured by sphygmomanometer while participant was in supine position. Conditions were kept constant from visit to visit including observer, participant's same arm, cuff size, supine position, location, temperature, noise level. The same size BP cuff which was properly sized and calibrated, was used to measure BP each time.
Time Frame: Baseline, Week 2, 4, 12, 24, 36, 48, 60, 72, 84, 96
Population: The safety analysis set included all participants in the FAS who received at least 1 dose of the study medication. Here, 'n' signifies participants evaluable for this outcome measure at given time points for each group.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 482 | 485 | 485
millimeters of mercury (mmHg)
  Baseline (n =482, 485, 485) | 127.04 (12.42) | 127.45 (12.18) | 127.45 (12.32)
  Change at Week 2 (n =459, 466, 462) | -0.06 (9.76) | 0.82 (10.66) | -0.01 (10.71)
  Change at Week 4 (n =467, 467, 465) | -1.08 (11.37) | 0.99 (11.12) | -0.94 (10.73)
  Change at Week 12 (n =450, 455, 461) | -0.11 (11.59) | 1.74 (12.09) | -0.76 (12.33)
  Change at Week 24 (n =425, 432, 439) | -0.47 (12.07) | 0.97 (12.14) | -0.73 (11.46)
  Change at Week 36 (n =385, 415, 418) | -0.11 (11.98) | -0.80 (12.02) | -1.58 (12.99)
  Change at Week 48 (n =377, 400, 410) | -0.83 (12.36) | -0.22 (11.39) | -0.28 (12.01)
  Change at Week 60 (n =360, 377, 384) | -1.02 (12.38) | 0.33 (12.02) | -1.36 (12.24)
  Change at Week 72 (n =357, 374, 370) | -0.82 (12.94) | -0.15 (13.00) | -0.20 (13.00)
  Change at Week 84 (n =346, 366, 362) | -1.43 (13.45) | -0.77 (12.98) | -1.15 (13.08)
  Change at Week 96 (n =344, 353, 356) | -0.55 (12.84) | 0.02 (12.52) | -0.71 (12.79)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 2; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis; LS mean difference = -0.27, 95% CI 2-sided [-1.50 to 0.96], Standard Error of Mean 0.63
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Superiority or Other; p = 0.326, Mixed Models Analysis; LS mean difference = 0.62, 95% CI 2-sided [-0.61 to 1.85], Standard Error of Mean 0.63
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 4; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.679, Mixed Models Analysis; LS mean difference = -0.27, 95% CI 2-sided [-1.56 to 1.01], Standard Error of Mean 0.66
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis; LS mean difference = 1.86, 95% CI 2-sided [0.57 to 3.14], Standard Error of Mean 0.66
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 12; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.399, Mixed Models Analysis; LS mean difference = 0.60, 95% CI 2-sided [-0.80 to 2.01], Standard Error of Mean 0.72
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = 2.52, 95% CI 2-sided [1.12 to 3.92], Standard Error of Mean 0.71
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 24; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis; LS mean difference = 0.30, 95% CI 2-sided [-1.08 to 1.68], Standard Error of Mean 0.70
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 7]; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; LS mean difference = 1.76, 95% CI 2-sided [0.39 to 3.13], Standard Error of Mean 0.70
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 36; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group x visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.109, Mixed Models Analysis; LS mean difference = 1.20, 95% CI 2-sided [-0.27 to 2.67], Standard Error of Mean 0.75
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; Week 36; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.163, Mixed Models Analysis; LS mean difference = 1.03, 95% CI 2-sided [-0.42 to 2.48], Standard Error of Mean 0.74
Statistical Analysis 11: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 48; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.424, Mixed Models Analysis; LS mean difference = -0.58, 95% CI 2-sided [-2.02 to 0.85], Standard Error of Mean 0.73
Statistical Analysis 12: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 11]; Test type: Superiority or Other; p = 0.635, Mixed Models Analysis; LS mean difference = 0.34, 95% CI 2-sided [-1.07 to 1.76], Standard Error of Mean 0.72
Statistical Analysis 13: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 60; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.855, Mixed Models Analysis; LS mean difference = 0.14, 95% CI 2-sided [-1.34 to 1.61], Standard Error of Mean 0.75
Statistical Analysis 14: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 13]; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis; LS mean difference = 1.84, 95% CI 2-sided [0.38 to 3.30], Standard Error of Mean 0.74
Statistical Analysis 15: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 72; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.292, Mixed Models Analysis; LS mean difference = -0.85, 95% CI 2-sided [-2.44 to 0.73], Standard Error of Mean 0.81
Statistical Analysis 16: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 15]; Test type: Superiority or Other; p = 0.897, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-1.47 to 1.68], Standard Error of Mean 0.80
Statistical Analysis 17: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 84; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis; LS mean difference = -0.72, 95% CI 2-sided [-2.36 to 0.92], Standard Error of Mean 0.84
Statistical Analysis 18: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 17]; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis; LS mean difference = 0.37, 95% CI 2-sided [-1.26 to 1.99], Standard Error of Mean 0.83
Statistical Analysis 19: Comparison: SD-0610 50 Milligram (mg) vs Placebo; Week 96; LS-Mean, 95 percent CI and P-values were obtained from a discrete time MMRM model with fixed effects for treatment group, visit, a treatment group*visit interaction, (collapsed) KLG, a (collapsed) KLG*visit interaction, baseline value, geographic region, gender, age and body mass index with an unstructured covariance matrix; Test type: Superiority or Other; p = 0.847, Mixed Models Analysis; LS mean difference = -0.16, 95% CI 2-sided [-1.73 to 1.42], Standard Error of Mean 0.80
Statistical Analysis 20: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 19]; Test type: Superiority or Other; p = 0.333, Mixed Models Analysis; LS mean difference = 0.77, 95% CI 2-sided [-0.79 to 2.34], Standard Error of Mean 0.80

43. Other Pre Specified Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 2, 4, 12, 24, 36, 48, 60, 72, 84 and 96
Description: BP was measured by sphygmomanometer while participant was in supine position. Conditions were kept constant from visit to visit including observer, participant's same arm, cuff size, supine position, location, temperature, noise level. The same size BP cuff which was properly sized and calibrated, was used to measure BP each time.
Time Frame: Baseline, Week 2, 4, 12, 24, 36, 48, 60, 72, 84, 96
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 482 | 485 | 485
mmHg
  Baseline (n =482, 485, 485) | 76.46 (7.68) | 77.06 (7.53) | 76.85 (7.71)
  Change at Week 2 (n =459, 466, 462) | 0.13 (6.63) | 0.58 (6.61) | 0.37 (7.07)
  Change at Week 4 (n =467, 467, 465) | 0.07 (7.04) | 0.78 (7.33) | -0.41 (7.11)
  Change at Week 12 (n =450, 455, 461) | 0.02 (7.29) | 1.21 (7.56) | 0.05 (7.58)
  Change at Week 24 (n =425, 432, 439) | 0.02 (7.46) | 0.53 (7.80) | -0.33 (7.52)
  Change at Week 36 (n =385, 415, 418) | -0.21 (7.86) | -0.31 (7.58) | -1.18 (7.86)
  Change at Week 48 (n =377, 400, 410) | -0.16 (8.28) | -0.19 (7.99) | -0.07 (7.67)
  Change at Week 60 (n =360, 377, 384) | -0.69 (7.56) | 0.10 (7.91) | -0.84 (8.32)
  Change at Week 72 (n =357, 374, 370) | -0.49 (8.06) | 0.30 (8.81) | -0.77 (8.14)
  Change at Week 84 (n= 346, 366, 362) | -0.39 (8.03) | -0.28 (7.93) | -0.78 (8.60)
  Change at Week 96 (n =344, 353, 356) | -0.21 (8.02) | -0.20 (8.82) | -0.70 (8.47)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Superiority or Other; p = 0.238, Mixed Models Analysis; LS mean difference = -0.49, 95% CI 2-sided [-1.31 to 0.32], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Superiority or Other; p = 0.815, Mixed Models Analysis; LS mean difference = 0.10, 95% CI 2-sided [-0.72 to 0.91], Standard Error of Mean 0.41
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Superiority or Other; p = 0.508, Mixed Models Analysis; LS mean difference = 0.28, 95% CI 2-sided [-0.54 to 1.10], Standard Error of Mean 0.42
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; LS mean difference = 1.20, 95% CI 2-sided [0.38 to 2.02], Standard Error of Mean 0.42
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Superiority or Other; p = 0.683, Mixed Models Analysis; LS mean difference = -0.18, 95% CI 2-sided [-1.07 to 0.70], Standard Error of Mean 0.45
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; LS mean difference = 1.21, 95% CI 2-sided [0.33 to 2.09], Standard Error of Mean 0.45
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 7]; Test type: Superiority or Other; p = 0.687, Mixed Models Analysis; LS mean difference = 0.18, 95% CI 2-sided [-0.71 to 1.07], Standard Error of Mean 0.45
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 7]; Test type: Superiority or Other; p = 0.050, Mixed Models Analysis; LS mean difference = 0.89, 95% CI 2-sided [-0.00 to 1.78], Standard Error of Mean 0.45
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 10]; Test type: Superiority or Other; p = 0.215, Mixed Models Analysis; LS mean difference = 0.60, 95% CI 2-sided [-0.35 to 1.54], Standard Error of Mean 0.48
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 10]; Test type: Superiority or Other; p = 0.042, Mixed Models Analysis; LS mean difference = 0.96, 95% CI 2-sided [0.03 to 1.89], Standard Error of Mean 0.47
Statistical Analysis 11: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 11]; Test type: Superiority or Other; p = 0.401, Mixed Models Analysis; LS mean difference = -0.42, 95% CI 2-sided [-1.41 to 0.56], Standard Error of Mean 0.50
Statistical Analysis 12: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 11]; Test type: Superiority or Other; p = 0.980, Mixed Models Analysis; LS mean difference = 0.01, 95% CI 2-sided [-0.96 to 0.99], Standard Error of Mean 0.50
Statistical Analysis 13: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 13]; Test type: Superiority or Other; p = 0.632, Mixed Models Analysis; LS mean difference = -0.24, 95% CI 2-sided [-1.25 to 0.76], Standard Error of Mean 0.51
Statistical Analysis 14: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 13]; Test type: Superiority or Other; p = 0.032, Mixed Models Analysis; LS mean difference = 1.08, 95% CI 2-sided [0.09 to 2.07], Standard Error of Mean 0.51
Statistical Analysis 15: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 15]; Test type: Superiority or Other; p = 0.668, Mixed Models Analysis; LS mean difference = -0.23, 95% CI 2-sided [-1.29 to 0.83], Standard Error of Mean 0.54
Statistical Analysis 16: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 15]; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; LS mean difference = 1.11, 95% CI 2-sided [0.06 to 2.16], Standard Error of Mean 0.54
Statistical Analysis 17: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 17]; Test type: Superiority or Other; p = 0.868, Mixed Models Analysis; LS mean difference = -0.09, 95% CI 2-sided [-1.13 to 0.95], Standard Error of Mean 0.53
Statistical Analysis 18: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 17]; Test type: Superiority or Other; p = 0.257, Mixed Models Analysis; LS mean difference = 0.59, 95% CI 2-sided [-0.43 to 1.62], Standard Error of Mean 0.52
Statistical Analysis 19: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 19]; Test type: Superiority or Other; p = 0.895, Mixed Models Analysis; LS mean difference = 0.07, 95% CI 2-sided [-1.00 to 1.15], Standard Error of Mean 0.55
Statistical Analysis 20: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 19]; Test type: Superiority or Other; p = 0.268, Mixed Models Analysis; LS mean difference = 0.60, 95% CI 2-sided [-0.46 to 1.67], Standard Error of Mean 0.54

44. Other Pre Specified Outcome: Change From Baseline in Heart Rate at Week 2, 4, 12, 24, 36, 48, 60, 72, 84 and 96
Time Frame: Baseline, Week 2, 4, 12, 24, 36, 48, 60, 72, 84, 96
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | SD-0610 50 Milligram (mg) | SD-0610 200 mg | Placebo
Number analyzed (Participants) | 482 | 485 | 485
beats per minute (bpm)
  Baseline (n =482, 485, 485) | 69.74 (9.11) | 69.12 (8.72) | 69.34 (8.26)
  Change at Week 2 (n =459, 466, 461) | 0.58 (7.35) | -0.29 (6.68) | 0.71 (7.55)
  Change at Week 4 (n =467, 466, 465) | 0.24 (7.53) | 0.23 (7.46) | 0.78 (7.77)
  Change at Week 12 (n =450, 455, 461) | 0.13 (7.70) | -0.17 (7.61) | 0.05 (8.24)
  Change at Week 24 (n =425, 432, 439) | 0.45 (8.30) | -0.42 (7.46) | 0.06 (8.37)
  Change at Week 36 (n =384, 415, 418) | -0.08 (8.58) | -0.07 (7.80) | 0.76 (8.41)
  Change at Week 48 (n =377, 399, 410) | -0.82 (8.45) | -1.37 (8.23) | -0.11 (8.59)
  Change at Week 60 (n =360, 377, 384) | -0.42 (8.37) | 0.04 (7.56) | 0.47 (8.90)
  Change at Week 72 (n =357, 374, 370) | -0.95 (8.75) | -0.99 (7.91) | 0.85 (9.56)
  Change at Week 84 (n =346, 366, 362) | -0.31 (8.65) | -0.15 (7.88) | 0.57 (8.64)
  Change at Week 96 (n =344, 353, 356) | -1.09 (8.91) | -0.61 (8.53) | 0.36 (8.61)
Statistical Analysis 1: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Superiority or Other; p = 0.908, Mixed Models Analysis; LS mean difference = -0.05, 95% CI 2-sided [-0.92 to 0.82], Standard Error of Mean 0.44
Statistical Analysis 2: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 1]; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis; LS mean difference = -1.18, 95% CI 2-sided [-2.05 to -0.31], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Superiority or Other; p = 0.440, Mixed Models Analysis; LS mean difference = -0.35, 95% CI 2-sided [-1.25 to 0.54], Standard Error of Mean 0.46
Statistical Analysis 4: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 3]; Test type: Superiority or Other; p = 0.140, Mixed Models Analysis; LS mean difference = -0.67, 95% CI 2-sided [-1.57 to 0.22], Standard Error of Mean 0.46
Statistical Analysis 5: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Superiority or Other; p = 0.474, Mixed Models Analysis; LS mean difference = 0.33, 95% CI 2-sided [-0.58 to 1.24], Standard Error of Mean 0.46
Statistical Analysis 6: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 5]; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis; LS mean difference = -0.41, 95% CI 2-sided [-1.32 to 0.50], Standard Error of Mean 0.46
Statistical Analysis 7: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 7]; Test type: Superiority or Other; p = 0.186, Mixed Models Analysis; LS mean difference = 0.66, 95% CI 2-sided [-0.32 to 1.64], Standard Error of Mean 0.50
Statistical Analysis 8: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 7]; Test type: Superiority or Other; p = 0.185, Mixed Models Analysis; LS mean difference = -0.66, 95% CI 2-sided [-1.63 to 0.32], Standard Error of Mean 0.50
Statistical Analysis 9: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 10]; Test type: Superiority or Other; p = 0.334, Mixed Models Analysis; LS mean difference = -0.51, 95% CI 2-sided [-1.53 to 0.52], Standard Error of Mean 0.52
Statistical Analysis 10: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 10]; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; LS mean difference = -0.99, 95% CI 2-sided [-2.00 to 0.02], Standard Error of Mean 0.52
Statistical Analysis 11: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 11]; Test type: Superiority or Other; p = 0.539, Mixed Models Analysis; LS mean difference = -0.33, 95% CI 2-sided [-1.38 to 0.72], Standard Error of Mean 0.54
Statistical Analysis 12: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 11]; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; LS mean difference = -1.26, 95% CI 2-sided [-2.30 to -0.22], Standard Error of Mean 0.53
Statistical Analysis 13: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 13]; Test type: Superiority or Other; p = 0.365, Mixed Models Analysis; LS mean difference = -0.48, 95% CI 2-sided [-1.52 to 0.56], Standard Error of Mean 0.53
Statistical Analysis 14: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 13]; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis; LS mean difference = -0.44, 95% CI 2-sided [-1.47 to 0.59], Standard Error of Mean 0.52
Statistical Analysis 15: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 15]; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; LS mean difference = -1.32, 95% CI 2-sided [-2.43 to -0.21], Standard Error of Mean 0.57
Statistical Analysis 16: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 15]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; LS mean difference = -1.87, 95% CI 2-sided [-2.98 to -0.77], Standard Error of Mean 0.56
Statistical Analysis 17: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 17]; Test type: Superiority or Other; p = 0.269, Mixed Models Analysis; LS mean difference = -0.60, 95% CI 2-sided [-1.66 to 0.46], Standard Error of Mean 0.54
Statistical Analysis 18: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 17]; Test type: Superiority or Other; p = 0.104, Mixed Models Analysis; LS mean difference = -0.87, 95% CI 2-sided [-1.92 to 0.18], Standard Error of Mean 0.54
Statistical Analysis 19: Comparison: SD-0610 50 Milligram (mg) vs Placebo; [analysis description as in outcome 42, analysis 19]; Test type: Superiority or Other; p = 0.038, Mixed Models Analysis; LS mean difference = -1.18, 95% CI 2-sided [-2.30 to -0.06], Standard Error of Mean 0.57
Statistical Analysis 20: Comparison: SD-0610 200 mg vs Placebo; [analysis description as in outcome 42, analysis 19]; Test type: Superiority or Other; p = 0.041, Mixed Models Analysis; LS mean difference = -1.16, 95% CI 2-sided [-2.28 to -0.05], Standard Error of Mean 0.57

ADVERSE EVENTS:
Time Frame: Baseline up to Week 111
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non serious in another participant, or one participant may have experienced both a serious and non serious event during the study.
Arm/Group | SD-6010 50 Milligram (mg) | SD-6010 200 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 43/482 | 61/485 | 49/485
Other Adverse Events (participants affected / at risk) | 365/482 | 371/485 | 360/485
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-6010 50 Milligram (mg) (N=482) | SD-6010 200 mg (N=485) | Placebo (N=485)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 3
Bradyarrhythmia (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 2
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 3 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1
Internal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 4 | 3 | 2
Device dislocation (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Medical device complication (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Gastric ulcer helicobacter (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Infectious peritonitis (Infections and infestations) | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Deep vein thrombosis postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 1 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1
Borrelia test positive (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0
Lacunar infarction (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Spinal vascular disorder (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 2
Tremor (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Bladder perforation (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urogenital disorder (Renal and urinary disorders) | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 3 | 0
Endometrial disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SD-6010 50 Milligram (mg) (N=482) | SD-6010 200 mg (N=485) | Placebo (N=485)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 9
Eosinophilia (Blood and lymphatic system disorders) | 1 | 1 | 2
Hypochromasia (Blood and lymphatic system disorders) | 0 | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 2 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 4
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 2 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 3 | 0
Bundle branch block left (Cardiac disorders) | 0 | 2 | 1
Bundle branch block right (Cardiac disorders) | 0 | 0 | 3
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 1 | 0 | 0
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 3 | 7 | 3
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 2 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 1 | 4
Brain malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0
Vascular anomaly (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 3 | 2 | 1
Ear disorder (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 4 | 1
Ear pruritus (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 1 | 3
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 7 | 4 | 7
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 1
Goitre (Endocrine disorders) | 4 | 1 | 4
Hypogonadism (Endocrine disorders) | 0 | 0 | 1
Hypoparathyroidism (Endocrine disorders) | 0 | 0 | 1
Thyroid cyst (Endocrine disorders) | 0 | 0 | 1
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 6 | 3 | 3
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1
Age-related macular degeneration (Eye disorders) | 0 | 1 | 0
Arcus lipoides (Eye disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 5 | 7 | 2
Cataract subcapsular (Eye disorders) | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 2 | 4 | 1
Dry eye (Eye disorders) | 2 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 1
Eye allergy (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 1
Eyelid irritation (Eye disorders) | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 1 | 1 | 0
Maculopathy (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Ocular hypertension (Eye disorders) | 1 | 0 | 0
Papilloedema (Eye disorders) | 0 | 1 | 0
Retinal detachment (Eye disorders) | 3 | 0 | 0
Retinal disorder (Eye disorders) | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 1 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 5 | 4 | 8
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 11 | 14
Abdominal pain lower (Gastrointestinal disorders) | 2 | 4 | 2
Abdominal pain upper (Gastrointestinal disorders) | 9 | 13 | 12
Abdominal tenderness (Gastrointestinal disorders) | 1 | 2 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 8 | 9 | 8
Dental caries (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 22 | 27 | 29
Diverticulum (Gastrointestinal disorders) | 2 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 10 | 14 | 14
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 5 | 2 | 4
Food poisoning (Gastrointestinal disorders) | 2 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 4 | 11 | 4
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 12 | 9
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gingival recession (Gastrointestinal disorders) | 0 | 1 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 6 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 2 | 2
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 20 | 15 | 14
Oesophageal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1
Omental infarction (Gastrointestinal disorders) | 1 | 0 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 2 | 0 | 1
Steatorrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Swollen tongue (Gastrointestinal disorders) | 1 | 0 | 0
Tooth impacted (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 5 | 2 | 8
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 9 | 12 | 3
Application site dermatitis (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 3 | 2 | 1
Chest discomfort (General disorders) | 0 | 2 | 1
Chest pain (General disorders) | 6 | 8 | 8
Chills (General disorders) | 1 | 0 | 1
Cyst (General disorders) | 1 | 0 | 1
Facial pain (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 10 | 12 | 13
Feeling cold (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 2 | 6 | 1
Injection site erythema (General disorders) | 1 | 0 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0
Irritability (General disorders) | 4 | 1 | 1
Malaise (General disorders) | 0 | 1 | 1
Medical device pain (General disorders) | 1 | 0 | 0
Medical device site reaction (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 1
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 15 | 15 | 19
Pain (General disorders) | 4 | 6 | 2
Polyp (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 2
Soft tissue inflammation (General disorders) | 0 | 0 | 1
Tenderness (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 0 | 2
Ulcer (General disorders) | 1 | 0 | 0
Ulcer haemorrhage (General disorders) | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 1 | 0
Biliary tract disorder (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 1 | 2
Gallbladder polyp (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 2 | 0 | 2
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 2
Sarcoidosis (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 1 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0
Acariasis (Infections and infestations) | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 5 | 6 | 5
Appendicitis (Infections and infestations) | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 1 | 0
Borrelia infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 25 | 30 | 20
Bronchitis viral (Infections and infestations) | 0 | 1 | 1
Candidiasis (Infections and infestations) | 3 | 2 | 0
Carbuncle (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 3 | 8 | 6
Cystitis (Infections and infestations) | 3 | 6 | 3
Device related infection (Infections and infestations) | 1 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 1 | 3
Ear infection (Infections and infestations) | 8 | 8 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 1
Erythema migrans (Infections and infestations) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 2 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 2 | 1
Fungal skin infection (Infections and infestations) | 0 | 2 | 0
Gastroenteritis (Infections and infestations) | 9 | 9 | 4
Gastroenteritis viral (Infections and infestations) | 5 | 3 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 1 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 1
Giardiasis (Infections and infestations) | 0 | 0 | 2
Gingival infection (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 1 | 1 | 1
Herpes ophthalmic (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 1 | 1
Herpes virus infection (Infections and infestations) | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 9 | 5 | 5
Hordeolum (Infections and infestations) | 0 | 1 | 0
Impetigo (Infections and infestations) | 0 | 1 | 0
Infected cyst (Infections and infestations) | 0 | 1 | 0
Infection parasitic (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 13 | 12 | 14
Labyrinthitis (Infections and infestations) | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 2 | 2
Laryngitis viral (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 3
Lyme disease (Infections and infestations) | 0 | 0 | 2
Mastitis bacterial (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 33 | 41 | 25
Onychomycosis (Infections and infestations) | 3 | 2 | 2
Oral candidiasis (Infections and infestations) | 0 | 2 | 0
Oral herpes (Infections and infestations) | 2 | 2 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 2 | 0 | 1
Otitis media (Infections and infestations) | 2 | 0 | 3
Otitis media acute (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 7 | 16 | 7
Pharyngitis bacterial (Infections and infestations) | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 4 | 2 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 6 | 4
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 1
Renal abscess (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0
Sinusitis (Infections and infestations) | 18 | 18 | 14
Skin infection (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 1
Tooth abscess (Infections and infestations) | 6 | 4 | 2
Tracheitis (Infections and infestations) | 0 | 0 | 1
Typhus (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 40 | 31 | 30
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 24 | 21 | 26
Vaginal infection (Infections and infestations) | 1 | 2 | 1
Viral infection (Infections and infestations) | 2 | 2 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1
Viral tonsillitis (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 2 | 2
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 1 | 0
Vulvovaginitis (Infections and infestations) | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 4 | 4 | 2
Animal bite (Injury, poisoning and procedural complications) | 1 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 3 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Bone fragmentation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 2 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 12 | 12 | 10
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 2 | 3 | 3
Eschar (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 4 | 4 | 5
Fall (Injury, poisoning and procedural complications) | 26 | 41 | 28
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 4 | 2
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Foreign body in eye (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 2 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 2 | 4 | 1
Laceration (Injury, poisoning and procedural complications) | 3 | 4 | 2
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 8 | 11 | 7
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 6 | 6 | 9
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 8 | 5 | 6
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 0 | 2
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 3
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Blood amylase increased (Investigations) | 3 | 6 | 3
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium increased (Investigations) | 3 | 2 | 0
Blood cholesterol abnormal (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 3 | 2
Blood creatine increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 2 | 3 | 4
Blood glucose increased (Investigations) | 2 | 3 | 3
Blood potassium decreased (Investigations) | 2 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 13 | 24 | 21
Blood testosterone decreased (Investigations) | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 4 | 0 | 0
Blood uric acid increased (Investigations) | 2 | 1 | 3
Blood urine present (Investigations) | 2 | 0 | 1
Body temperature increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 3 | 1 | 0
Ceruloplasmin increased (Investigations) | 0 | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 1 | 0 | 0
Eosinophil count increased (Investigations) | 1 | 1 | 0
Femoral bruit (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 10 | 4
Haematocrit decreased (Investigations) | 1 | 0 | 1
Haematology test abnormal (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Heart rate increased (Investigations) | 0 | 0 | 1
Heart rate irregular (Investigations) | 0 | 1 | 0
Helicobacter test positive (Investigations) | 1 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 2 | 0
Lipase increased (Investigations) | 7 | 8 | 7
Liver function test abnormal (Investigations) | 3 | 1 | 3
Low density lipoprotein increased (Investigations) | 1 | 0 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 1
Pancreatic enzymes increased (Investigations) | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 2 | 1
Protein urine present (Investigations) | 1 | 0 | 0
Red blood cell burr cells present (Investigations) | 0 | 1 | 0
Serum ferritin increased (Investigations) | 0 | 0 | 1
Tandem gait test abnormal (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 2 | 2
Ultrasound kidney abnormal (Investigations) | 0 | 1 | 0
Vitamin B12 decreased (Investigations) | 0 | 0 | 1
Vitamin D decreased (Investigations) | 2 | 0 | 0
Waist circumference increased (Investigations) | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 1
Weight increased (Investigations) | 1 | 7 | 5
White blood cell count abnormal (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0
Cholesterosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 4 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 3 | 5
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 9 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 4
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 6 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 2 | 5
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 69 | 65 | 65
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 8 | 4
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Articular calcification (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 31 | 32 | 43
Bone loss (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 12 | 2 | 7
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Joint lock (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 14 | 8 | 7
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lordosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 9 | 3
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 13 | 17
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 5
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 12 | 7
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 21 | 23 | 14
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 19 | 21
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 9
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Resorption bone increased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 6 | 5
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3
Spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 3 | 2 | 4
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 9 | 14 | 11
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Morton's neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Paranasal sinus benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 1 | 0 | 2
Carotid artery disease (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 3 | 2 | 6
Cerebral microangiopathy (Nervous system disorders) | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0
Cluster headache (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 17 | 22 | 11
Dysgeusia (Nervous system disorders) | 3 | 1 | 1
Headache (Nervous system disorders) | 32 | 27 | 18
Hemiparesis (Nervous system disorders) | 1 | 2 | 0
Hypertonia (Nervous system disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 4 | 5 | 2
Hyporeflexia (Nervous system disorders) | 0 | 0 | 1
Lethargy (Nervous system disorders) | 3 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 2 | 0 | 2
Memory impairment (Nervous system disorders) | 1 | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 6 | 7 | 1
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Multiple sclerosis (Nervous system disorders) | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 1
Nerve compression (Nervous system disorders) | 2 | 0 | 3
Neuralgia (Nervous system disorders) | 1 | 0 | 1
Neuritis (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 2
Paraesthesia (Nervous system disorders) | 5 | 3 | 3
Parkinson's disease (Nervous system disorders) | 1 | 2 | 1
Presyncope (Nervous system disorders) | 1 | 1 | 0
Radicular syndrome (Nervous system disorders) | 1 | 0 | 0
Radiculitis (Nervous system disorders) | 1 | 0 | 1
Radiculitis cervical (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 3 | 2 | 0
Sciatic nerve neuropathy (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 4 | 10 | 2
Sinus headache (Nervous system disorders) | 1 | 3 | 1
Sleep phase rhythm disturbance (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 2
Syncope (Nervous system disorders) | 3 | 1 | 1
Tension headache (Nervous system disorders) | 0 | 2 | 1
Tremor (Nervous system disorders) | 2 | 2 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1
Vascular encephalopathy (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 6 | 7 | 5
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 12 | 12 | 6
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Emotional distress (Psychiatric disorders) | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 9 | 5 | 7
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 5 | 0 | 1
Haematuria (Renal and urinary disorders) | 5 | 2 | 6
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 4 | 3
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 3 | 0
Renal cyst (Renal and urinary disorders) | 2 | 1 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 2 | 1 | 1
Urethral disorder (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 2 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 1 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 1
Breast cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 1 | 1 | 2
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0
Erection increased (Reproductive system and breast disorders) | 0 | 1 | 0
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Menopausal disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 2 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 1 | 0
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 1 | 0
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 3
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 8
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 2
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 5
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3
Rhinitis perennial (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Cutis laxa (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 3 | 8
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 2 | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2 | 4
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 5
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 12 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 3 | 4
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Bleeding varicose vein (Vascular disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2
Diastolic hypertension (Vascular disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 3 | 1 | 0
Haematoma (Vascular disorders) | 2 | 1 | 2
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 2 | 1 | 4
Hypertension (Vascular disorders) | 34 | 27 | 19
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 3 | 0 | 3
Phlebitis deep (Vascular disorders) | 1 | 0 | 0
Phlebitis superficial (Vascular disorders) | 0 | 0 | 1
Systolic hypertension (Vascular disorders) | 0 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 3 | 0
Venous insufficiency (Vascular disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.